CLINICAL TRIAL: NCT02367794
Title: A Phase III, Open-Label, Multicenter, Randomized Study Evaluating the Efficacy and Safety of Atezolizumab (MPDL3280A, Anti-PD-L1 Antibody) in Combination With Carboplatin+Paclitaxel or Atezolizumab in Combination With Carboplatin+Nab-Paclitaxel Versus Carboplatin+Nab-Paclitaxel in Chemotherapy-Naive Patients With Stage IV Squamous Non-Small Cell Lung Cancer
Brief Title: A Study of Atezolizumab in Combination With Carboplatin + Paclitaxel or Carboplatin + Nab-Paclitaxel Compared With Carboplatin + Nab-Paclitaxel in Participants With Stage IV Squamous Non-Small Cell Lung Cancer (NSCLC) [IMpower131]
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29437; 2014-003208-59 (EudraCT Number)
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — atezolizumab; Antibodies; Carboplatin; 130-nm albumin-bound paclitaxel; Paclitaxel

ARMS (3):
- Arm A: Atezolizumab + Paclitaxel + Carboplatin (Experimental): The induction phase of the study will consist of four or six cycles; atezolizumab, paclitaxel, and carboplatin will be administered on Day 1 of each 21-day cycle. The Day 1 order of drug administration is as follows: atezolizumab, then paclitaxel, then carboplatin. Participants who experience no further clinical benefit at any time during the induction phase will discontinue all study treatments. In the absence of the above criteria, after the 4- or 6-cycle induction phase, participants will begin maintenance therapy with atezolizumab. Atezolizumab will be continued as long as there is a clinical benefit to the participant.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-programmed death-ligand 1 (anti-PD-L1) antibody; Drug: Carboplatin; Drug: Paclitaxel
- Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin (Experimental): The induction phase of the study will consist of four or six cycles; atezolizumab and carboplatin will be administered on Day 1 of each 21-day cycle. Nab-Paclitaxel will be administered on Days 1, 8, and 15 of each 21-day cycle. The Day 1 order of drug administration is as follows: atezolizumab, then nab-paclitaxel, then carboplatin. Participants who experience no further clinical benefit at any time during the induction phase will discontinue all study treatments. In the absence of the above criteria, after the 4- or 6-cycle induction phase, participants will begin maintenance therapy with atezolizumab. Atezolizumab will be continued as long as there is a clinical benefit to the participant.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-programmed death-ligand 1 (anti-PD-L1) antibody; Drug: Carboplatin; Drug: Nab-Paclitaxel
- Arm C: Nab-Paclitaxel + Carboplatin (Active Comparator): The induction phase of the study will consist of four or six cycles; carboplatin will be administered on Day 1 of each 21-day cycle, nab-paclitaxel will be administered on Days 1, 8, and 15 of each 21-day cycle. The Day 1 order of drug administration is as follows: nab-paclitaxel, then carboplatin. Participants who experience disease progression at any time during the induction phase will discontinue all study treatment. In the maintenance phase, participants will receive best supportive care.
  Interventions: Drug: Carboplatin; Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A), an engineered anti-programmed death-ligand 1 (anti-PD-L1) antibody — Atezolizumab 1200 milligrams (mg) intravenous infusion (IV) on day 1 of each 21-day cycle.
  Other Names: Tecentriq
  Arms: Arm A: Atezolizumab + Paclitaxel + Carboplatin; Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin
Drug: Carboplatin — Carboplatin area under the concentration curve (AUC) 6 milligrams per milliliter per minute (mg/mL/min) on Day 1 of each 21-day cycle for 4 or 6 cycles.
Drug: Nab-Paclitaxel — Nab-paclitaxel 100 milligrams per meter squared (mg/m^2) IV on Day 1, 8, and 15 of each 21-day cycle for 4 or 6 cycles.
  Arms: Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin; Arm C: Nab-Paclitaxel + Carboplatin
Drug: Paclitaxel — Paclitaxel 200 mg/m^2 IV on Day 1 of each 21-day cycle for 4 or 6 cycles. Participants of Asian race/ethnicity will be administered paclitaxel 175 mg/m^2 IV.
  Arms: Arm A: Atezolizumab + Paclitaxel + Carboplatin

SUMMARY:
This randomized, open-label study will evaluate the safety and efficacy of atezolizumab (MPDL3280A) in combination with carboplatin + paclitaxel or carboplatin + nab-paclitaxel compared with treatment with carboplatin + nab-paclitaxel in chemotherapy-naive participants with Stage IV squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Histologically or cytologically confirmed, treatment-naïve Stage IV squamous NSCLC
* Previously obtained archival tumor tissue or tissue obtained from biopsy at screening
* Measurable disease as defined by RECIST v1.1
* Adequate hematologic and end organ function

Exclusion Criteria:

* Active or untreated central nervous system (CNS) metastasis
* Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome
* Pregnant or lactating women
* History of autoimmune disease
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest Computed Tomography (CT) scan, History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Positive test for Human Immunodeficiency Virus (HIV)
* Active hepatitis B or hepatitis C
* Prior treatment with cluster of differentiation 137 (CD137) agonists or immune checkpoint blockade therapies, anti-programmed death-1 (anti-PD-1), and anti-PD-L1 therapeutic antibody
* Severe infection within 4 weeks prior to randomization
* Significant history of cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1021 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2021-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (242):
- United States (57):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - Southern CA Permanente Med Grp, Bellflower, California
  - Kaiser Permanente Oakland Medical Center, Oakland, California
  - Kaiser Permanente - Sacramento Medical Center and Medical Offices, Sacramento, California
  - Kaiser Permanente - San Leandro Medical Center, San Leandro, California
  - Kaiser Permanente - Santa Clara, Santa Clara, California
  - Kaiser Permanente; Oncology Clinical Trials, Vallejo, California
  - Kaiser Permanente - Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Holy Cross Hospital Inc, Fort Lauderdale, Florida
  - SCRI Florida Cancer Specialists South, Fort Myers, Florida
  - Florida Cancer Specialists, Palm Beach Gardens, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Florida Cancer Specialists (St. Petersburg - St. Anthony's Professional Building), St. Petersburg, Florida
  - University Cancer & Blood Center, LLC; Research, Athens, Georgia
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital, Carrollton, Georgia
  - Central Georgia Cancer Care PC, Macon, Georgia
  - Southeastern Regional Medical Center, Inc., Newnan, Georgia
  - University of Chicago, Chicago, Illinois
  - Joliet Oncology-Hematology; Associates, Ltd., Joliet, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Fort Wayne Med Oncology & Hematology Inc, Fort Wayne, Indiana
  - Hematology-Oncology; Associates of the Quad Cities, Bettendorf, Iowa
  - Siouxland Hematology/Oncology, Sioux City, Iowa
  - Lahey Clinic Med Ctr, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - New England Cancer Specialists, Scarborough, Maine
  - Southcoast Health System; Southcoast Centers For Cancer Care, Fairhaven, Massachusetts
  - St. Joseph Mercy Health System, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - St. Luke's Regional Cancer Center, Duluth, Minnesota
  - Hematology and Oncology Associates at Bridgepoint, Tupelo, Mississippi
  - Billings Clinic, Billings, Montana
  - Valley Hospital; Oncology Research, Paramus, New Jersey
  - Regional Cancer Care Associates LLC, Sewell, New Jersey
  - Clinical Research Alliance, Westbury, New York
  - W.G. Bill Hefner VA Medical Center, Salisbury, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Mark H. Zangmeister Center, Columbus, Ohio
  - Oncology Hematology Care, Inc., Hamilton, Ohio
  - Oregon Health & Science Uni, Portland, Oregon
  - St. Luke's Cancer Care Associates, Bethlehem, Pennsylvania
  - Maryland Oncology Hematology (Lanham) - USOR, Gettysburg, Pennsylvania
  - Allegheny Cancer Center, Pittsburgh, Pennsylvania
  - Univ of Pittsburgh Medical Ctr, Pittsburgh, Pennsylvania
  - SCRI Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - SCRI The Center For Cancer and Blood Disorders, Denton, Texas
  - Longview Cancer Center, Longview, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - Providence Regional Cancer Partnership, Everett, Washington
  - Medical Oncology Associates, Spokane, Washington
- Argentina (6):
  - Fundación CENIT para la Investigación en Neurociencias, Buenos Aires
  - Sanatorio Allende, Córdoba
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - Clínica Pergamino, Pergamino
  - Fundacion Koriza, Santa Rosa
  - Centro de Investigacion; Clinica - Clinica Viedma S.A., Viedma
- Australia (10):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Calvary Mater Newcastle; Medical Oncology, Waratah, New South Wales
  - Prince Charles Hospital, Chermside, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Austin Health, Heidelberg, Victoria
  - Cabrini Hospital Malvern, Malvern, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Paracelsus Medizinische Privatuniversität, Salzburg, Austria
- Belgium (5):
  - Cliniques Universitaires St-Luc, Brussels
  - CHU Sart-Tilman, Liège
  - Clinique Ste-Elisabeth, Namur
  - Werken Glorieux VZW, Ronse
  - GasthuisZusters Antwerpen, Wilrijk
- Brazil (10):
  - Cenantron - Centro Avancado de Tratamento Oncologico, Belo Horizonte, Minas Gerais
  - Instituto Do Cancer Delondrina_X; Unidade De Pesquisa Clinica, Londrina, Paraná
  - Liga Norte Riograndense Contra O Câncer, Natal, Rio Grande do Norte
  - IPCEM; Instituto de Pesquisa de Estudos Multicêntricos, Caxias do Sul, Rio Grande do Sul
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - *X*Fundação Pio XII Hospital de Câncer de Barretos, Barretos, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Do Cancer A C Camargo, São Paulo, São Paulo
- Bulgaria (2):
  - Multiprofile Hospital for Active Treatment Central Onco Hospital OOD, Plovdiv
  - Multiprofile Hospital for Active Treatment Serdika EOOD, Sofia
- Canada (6):
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - William Osler Health Centre, Etobicoke, Ontario
  - Lakeridge Health Center, Oshawa, Ontario
  - Cite de La Sante de Laval; Hemato-Oncologie, Laval, Quebec
  - Hôpital du Sacré-Coeur de Montreal, Montreal, Quebec
  - St. Jerome Medical Research, Saint-Jérôme, Quebec
- Chile (2):
  - Health & Care SPA, Santiago
  - Sociedad de Investigaciones Medicas Ltda (SIM), Temuco
- France (10):
  - CHU de Grenoble, Grenoble
  - Ctr Jean Bernard Clin V. Hugo; Service d'Oncologie Méd, Le Mans
  - Centre Léon Bérard Centre Régional de Lutte Contre Le Cancer Rhône Alpes, Lyon
  - Clinique Clémentville, Montpellier
  - Hopital de La Source, Orléans
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital de Pontchaillou; Service de Pneumologie, Rennes
  - Centre Hospitalier Regional Sud Reunion; Service de Pneumologie, Saint-Pierre
  - CH de Saint Quentin, Saint-Quentin
  - Hôpital d'Instruction des Armées de Sainte Anne; Service Pharmacie Essais Cliniques, Toulon
- Germany (20):
  - Charite - Universitätsmedizin Berlin, Berlin
  - Ev.Krankenhaus Bielefeld gGmbH; Klinik für Innere Medizin und Geriatrie, Bielefeld
  - Augusta Kranken-Anstalt gGmbH, Bochum
  - Kliniken der Stadt Koln gGmbH, Cologne
  - Universitätsklinikum "Carl Gustav Carus" der Technischen Universität Dresden, Dresden
  - St. Elisabethen Krankenhaus, Frankfurt am Main
  - Robert Bosch Krankenhaus; Pneumologie und pneumologische Onkologie, Gerlingen
  - LungenClinic Großhansdorf GmbH, Großhansdorf
  - Krankenhaus Martha-Maria; Halle-Dolau gGmbH, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Harburg, Hamburg
  - Lungenklinik Hemer, Hemer
  - Universität Des Saarlandes; Klinik für Innere Medizin V, Homburg
  - Fachklinik für Lungenerkrankungen, Immenhausen
  - Johannes Wesling Klinikum Minden; Hämatologie, Onkologie, Hämostaseologie und Palliativmedizin, Minden
  - Klinikum Bogenhausen; Klinik für Pneumologie und Pneumologische Onkologie, München
  - Krankenhaus Barmherzige Bruder Regensburg, Regensburg
  - Klinikum der Universität Regensburg, Regensburg
  - Stiftung Mathias-Spital Rheine, Rheine
  - Schwarzwald-Baar Klinikum/VS GmbH; Onkologie/Hämatologie/Infektologie, Villingen-Schwenningen
- Israel (7):
  - Soroka Medical Center, Beersheba
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Meir Medical Center; Oncology, Kfar Saba
  - Rabin Medical Center, Petach Tiqwa
  - Chaim Sheba Medical Center; Oncology Dept, Ramat Gan
  - Rambam Health Corporation; Oncology Institute, Rambam
  - Tel Aviv Sourasky Medical Ctr; Oncology, Tel Aviv
- Italy (12):
  - IRCCS Giovanni Paolo II Istituto Oncologico, Bari, Apulia
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specialita San Giuseppe Moscati, Avellino, Campania
  - AORN A Cardarelli, Napoli, Campania
  - Azienda Ospedaliero Universitaria Seconda Università degli Studi di Napoli; Farmacia Centralizzata, Napoli, Campania
  - Istituto Nazionale per lo Studio e la Cura dei Tumori Fondazione G. Pascale, Napoli, Campania
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - ASL 3 Genovese; DSM, Genoa, Liguria
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy
  - Policlinico Vittorio Emanuele, Catania, Sicily
  - Ospedale Civile - Livorno, Livorno, Tuscany
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Ospedale Silvestrini, Perugia, Umbria
- Japan (24):
  - Aichi Cancer Center Hospital; Respiratory Medicine, Aichi
  - Nagoya University Hospital; Respiratory Medicine, Aichi
  - National Cancer Center Hospital East; Thoracic Oncology, Chiba
  - National Hospital Organization Shikoku Cancer Center; Internal Medicine, Ehime
  - National Hospital Organization Kyushu Medical Center; Respiratory Internal Medicine, Fukuoka
  - Kyushu University Hospital; Respiratory, Fukuoka
  - Kobe City Medical Center General Hospital; Respiratory Medicine, Hyōgo
  - National Hospital Organization Himeji Medical Center, Hyōgo
  - Hyogo Cancer Center; Thoracic Oncology, Hyōgo
  - Ibaraki Prefectural Central Hospital; Division of respiratory, Ibaraki
  - Kanagawa Cancer Center;Thoracic Oncology, Kanagawa
  - Kyoto University Hospital, Respiratory Medicine, Kyoto
  - Sendai Kousei Hospital; Pulmonary Medicine, Miyagi
  - Niigata University Medical & Dental Hospital; Respiratory Medicine and Infectious Disease, Niigata
  - Okayama University Hospital; Respiratory and Allergy Medicine, Okayama
  - Osaka International Cancer Institute; Thoracic Oncology, Osaka
  - Osaka City Uni Hospital; Respiratory Medicine, Osaka
  - Kansai Medical university Hospital; Thoracic Oncology, Osaka
  - Osaka Habikino Medical Center, Osaka
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakaishi
  - Saitama Cancer Center; Thoracic Oncology, Satima
  - Shizuoka Cancer Center; Thoracic Oncology, Shizuoka
  - National Cancer Center Hospital; Thoracic Medical Oncology, Tokyo
  - Tokyo Medical University Hospital; Dept of Surgery, Tokyo
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga East Clinical University Hospital Latvian Oncology Centre, Riga
- National Cancer Institute, Vilnius, Lithuania
- Mexico (2):
  - Centro Universitario Contra El Cancer, Monterrey
  - Cancerología, Querétaro
- Netherlands (5):
  - VU Medisch Centrum; VU University Medical Center, Amsterdam
  - Het Nederlands Kanker Instituut Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Hospital; Afdeling Longgeneeskunde en Tuberculose, Eindhoven
  - St. Antonius Ziekenhuis; R&D Long, Nieuwegein
- Peru (3):
  - Centro Medico Monte Carmelo, Arequipa
  - Hospital Nacional Guillermo Almenara Irigoyen ESSALUD, Lima
  - Instituto Regional de Enfermedades Neoplásicas Del Norte, Trujillo
- Portugal (5):
  - IPO de Lisboa; Servico de Pneumologia, Lisbon
  - Hospital Pulido Valente; Servico de Pneumologia, Lisbon
  - Centro Hospitalar do Porto - Hospital de Santo António, Porto
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil Epe, Porto
  - Hospital de Sao Joao; Servico de Pneumologia, Porto
- Russia (5):
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - Russian Oncology Research Center n.a. N.N. Blokhin, Moscow
  - Clinical Oncology Dispensary, Omsk
  - City Clinical Oncology Dispensary, Saint Petersburg
  - Volgograd Regional Clinical Oncology Dispensary, Volgograd
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
- Slovakia (3):
  - Univerzitna nemocnica Bratislava, Bratislava
  - Narodny onkologicky ustav, Bratislava
  - POKO Poprad s.r.o., Poprad
- Spain (24):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Instituto Catalan de Oncologia de Hospitalet (ICO); Servicio de Farmacia, L'Hospitalet de Llobregat, Barcelona
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla; Servicio de Oncologia, Santander, Cantabria
  - Complejo Hospitalario Universitario A Coruña, A Coruña, LA Coruña
  - Complejo Hospitalario Universitario Insular-Materno Infantil, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Nuestra Senora de Valme, Seville, Sevilla
  - Hospital Universitario de Canarias, S. Cristobal de La Laguna, Tenerife
  - Hospital del Mar, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Oncologia, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Lucus Augusti; Servicio de Oncologia, Lugo
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Fundación Jimenez Díaz, Madrid
  - Hospital Clinico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - HOSPITAL DE MADRID NORTE SANCHINARRO- CENTRO INTEGRAL ONCOLOGICO CLARA CAMPAL; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (7):
  - Changhua Christian Hospital; Hematology-Oncology, Changhua
  - Kaohsiung Medical University Hospital; Department of Urology, Kaohsiung City
  - Chi Mei Medical Center Liou Ying Campus, Liuying Township
  - Chang Gung Memorial Hospital Chiayi, Putzu
  - China Medical University Hospital, Taichung
  - National Taiwan Uni Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
- Ukraine (11):
  - Municipal Institution City Clinical Hospital #4 of Dnipro City Council - PPDS; Dept of Chemotherapy, Dnipropetrovsk, Katerynoslav Governorate
  - Uzhgorod Central City Clinical Hospital, Uzhhorod, Katerynoslav Governorate
  - MNPE Zaporizhzhia Regional Antitumor Center ZRC, Zaporizhzhia, Katerynoslav Governorate
  - Communal Non profit Enterprise Regional Center of Oncology; Oncosurgical dept of thoracic organs, Kharkiv, Kharkiv Governorate
  - Communal Nonprofit Enterprise Podilsky Regional Center Of Oncology OfTheVinnytsia Regional Council, Vinnytsia, KIEV Governorate
  - MI of the Lviv Regional Council Lviv Oncology Regional Treatment and Diagnostic Centre; Chemotherapy, Lviv, Volhynian Governorate
  - Municipal Institution Chernivtsi Regional Clinical Oncology Dispensary; Surgery Department #1, Chernivtsi
  - SI Institute of Medical Radiology n.a. S.P. Hryhoriev of NAMS of Ukraine, Kharkiv
  - ME Kryviy Rih Oncology Dispensary of Dnipropetrovs'k Regional Council; Chemotherapy Department, Kryvyi Rih
  - Poltava Regional Clinical Oncology Dispensary of Poltava Regional Council; Thoracic department, Poltava
  - Regional Municipal Institution Sumy Regional Clinical Oncology Dispensary, Sumy

REFERENCES:
- [Derived] Ton TGN, Pal N, Trinh H, Mahrus S, Bretscher MT, Machado RJM, Sadetsky N, Chaudhary N, Lu MW, Riely GJ. Replication of Overall Survival, Progression-Free Survival, and Overall Response in Chemotherapy Arms of Non-Small Cell Lung Cancer Trials Using Real-World Data. Clin Cancer Res. 2022 Jul 1;28(13):2844-2853. doi: 10.1158/1078-0432.CCR-22-0471. PMID 35511917

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 'Study Terminated By Sponsor' Reason for Not Completed is a data entry error; reason for not completed is unknown. The study was Completed and not Terminated.
Groups:
- Arm C: Nab-Paclitaxel + Carboplatin: The induction phase of the study consisted of four or six cycles; carboplatin was administered on Day 1 of each 21-day cycle, nab-paclitaxel was administered on Days 1, 8, and 15 of each 21-day cycle. The Day 1 order of drug administration was as follows: nab-paclitaxel, then carboplatin. Participants who experienced disease progression at any time during the induction phase discontinued all study treatment. In the maintenance phase, participants received best supportive care.
- Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin: The induction phase of the study consisted of four or six cycles; atezolizumab and carboplatin were administered on Day 1 of each 21-day cycle. Nab-Paclitaxel was administered on Days 1, 8, and 15 of each 21-day cycle. The Day 1 order of drug administration was as follows: atezolizumab, then nab-paclitaxel, then carboplatin. Participants who experienced no further clinical benefit at any time during the induction phase discontinued all study treatments. In the absence of the above criteria, after the 4- or 6-cycle induction phase, participants began maintenance therapy with atezolizumab. Atezolizumab was continued as long as there was clinical benefit to the participant.
- Arm A: Atezolizumab + Paclitaxel + Carboplatin: The induction phase of the study consisted of four or six cycles; atezolizumab, paclitaxel, and carboplatin were administered on Day 1 of each 21-day cycle. The Day 1 order of drug administration was as follows: atezolizumab, then paclitaxel, then carboplatin. Participants who experienced no further clinical benefit at any time during the induction phase discontinued all study treatments. In the absence of the above criteria, after the 4- or 6-cycle induction phase, participants began maintenance therapy with atezolizumab. Atezolizumab was continued as long as there was clinical benefit to the participant.
Period: Overall Study
Arm/Group | Arm C: Nab-Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Started | 340 | 343 | 338
Completed | 0 | 0 | 0
Not Completed | 340 | 343 | 338
Not completed — Death | 252 | 245 | 243
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Physician Decision | 0 | 5 | 3
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Withdrawal by Subject | 25 | 12 | 20
Not completed — Brain metastasis | 1 | 0 | 0
Not completed — Randomized in error | 0 | 0 | 1
Not completed — Patient unable to receive carboplatin | 0 | 0 | 1
Not completed — Hypercalcemia prior to C1D1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Study Terminated By Sponsor | 0 | 1 | 1
Not completed — Moved to Roll-Over Study | 0 | 15 | 13
Not completed — Sponsor Request | 60 | 57 | 45
Not completed — Moved into PTAP Study | 0 | 2 | 3
Not completed — Moved to Commercial Atezolizumab Use | 0 | 2 | 1
Not completed — Investigational Product Availability in Commercial Stock | 0 | 1 | 0
Not completed — Participant Enrolled in Extended Protocol | 0 | 1 | 0
Not completed — Discontinuation Matched Treatment Discontinuation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm C: Nab-Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin | Total
Number analyzed (Participants) | 340 | 343 | 338 | 1021
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.9 (8.1) | 64.0 (9.2) | 65.0 (8.3) | 64.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 63 | 60 | 186
  Male | 277 | 280 | 278 | 835
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 27 | 28 | 79
  Not Hispanic or Latino | 299 | 306 | 297 | 902
  Unknown or Not Reported | 17 | 10 | 13 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 3 | 5
  Asian | 37 | 41 | 34 | 112
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 7 | 4 | 3 | 14
  White | 290 | 289 | 290 | 869
  More than one race | 1 | 6 | 1 | 8
  Unknown or Not Reported | 4 | 2 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Determined by the Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) in the Intent-to-Treat (ITT) Population
Description: PFS is defined as the time between the date of randomization and the date of first documented disease progression or death, whichever occurs first, in the ITT population.
Time Frame: Up to approximately 30 months after first participant enrolled
Population: Intent To Treat (ITT) was defined as all randomized participants, irrespective of whether the assigned treatment was actually received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm C: Nab-Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 340 | 343 | 338
Months | 5.6 [5.5 to 5.7] | 6.5 [5.7 to 7.1] | 5.6 [5.5 to 6.9]
Statistical Analysis 1: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin; Test type: Superiority; p = 0.0006, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.64 to 0.88]

2. Primary Outcome: Overall Survival (OS) in the ITT Population
Description: OS is defined as the time between the date of randomization and date of death from any cause in the ITT population.
Time Frame: Up to approximately 39 months after first participant enrolled
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm C: Nab-Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 340 | 343 | 338
Months | 13.5 [12.2 to 15.1] | 14.2 [12.3 to 16.8] | 12.6 [11.6 to 14.7]
Statistical Analysis 1: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin; Test type: Superiority; p = 0.1581, Log Rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.73 to 1.05]

3. Secondary Outcome: OS in the in the Teff Population
Description: OS is defined as the time between the date of randomization and date of death from any cause in the in the Teff Population.
Time Frame: Up to approximately 39 months after first participant enrolled
Population: The Teff (>=-1.91) population and the Teff (<-1.91) population, defined as patients in the ITT population with Teff signature expression >=-1.91 and <-1.91, respectively.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Arm C: Nab-Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 322 | 313 | 308
Month
  Teff >=-1.91: number analyzed (Participants) | 147 | 124 | 123
  Teff >=-1.91 | 16.4 [12.2 to 19.7] | 17.4 [12.3 to 23.8] | 15.2 [13.4 to 22.8]
  Teff<-1.91: number analyzed (Participants) | 175 | 189 | 185
  Teff<-1.91 | 12.4 [11.2 to 14.3] | 13.0 [11.4 to 14.8] | 10.5 [9.1 to 12.6]
Statistical Analysis 1: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin; Teff >=-1.91 in ITT; Test type: Superiority — Stratified Analysis; p = 0.4451, Log Rank; Hazard Ratio (HR) = 0.876, 95% CI 2-sided [0.623 to 1.231]
Statistical Analysis 2: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm A: Atezolizumab + Paclitaxel + Carboplatin; Teff >=-1.91 in ITT; Test type: Superiority — Stratified Analysis; p = 0.7343, Log Rank; Hazard Ratio (HR) = 0.941, 95% CI 2-sided [0.664 to 1.335]
Statistical Analysis 3: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin; Teff <-1.91 Negative in ITT; Test type: Superiority — Stratified Analysis; p = 0.6610, Log Rank; Hazard Ratio (HR) = 0.942, 95% CI 2-sided [0.720 to 1.232]
Statistical Analysis 4: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm A: Atezolizumab + Paclitaxel + Carboplatin; Teff <-1.91 Negative in ITT; Test type: Superiority — Stratified Analysis; p = 0.0893, Log Rank; Hazard Ratio (HR) = 1.253, 95% CI 2-sided [0.965 to 1.627]

4. Secondary Outcome: PFS as Determined by the Investigator Using RECIST v1.1 in the Teff Population
Description: PFS is defined as the time between the date of randomization and the date of first documented disease progression or death, whichever occurs first, in the Teff Population.
Time Frame: Up to approximately 30 months after first participant enrolled
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm C: Nab-Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 322 | 313 | 308
Months
  Teff >=-1.91: number analyzed (Participants) | 147 | 124 | 123
  Teff >=-1.91 | 5.6 [5.1 to 5.7] | 7.0 [5.5 to 8.5] | 7.0 [5.6 to 9.7]
  Teff<-1.91: number analyzed (Participants) | 175 | 189 | 185
  Teff<-1.91 | 5.7 [5.5 to 6.6] | 6.2 [5.6 to 7.0] | 5.5 [4.5 to 5.6]
Statistical Analysis 1: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin; Teff>=-1.91; Test type: Superiority — Stratified Analysis; p = 0.0006, Log Rank; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.46 to 0.81]
Statistical Analysis 2: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm A: Atezolizumab + Paclitaxel + Carboplatin; Teff>=-1.91; Test type: Superiority — Stratified Analysis; p = 0.630, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.84 to 1.33]
Statistical Analysis 3: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin; Teff<-1.91; Test type: Superiority — Stratified Analysis; p = 0.258, Log Rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.70 to 1.10]
Statistical Analysis 4: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm A: Atezolizumab + Paclitaxel + Carboplatin; Teff<-1.91; Test type: Superiority — Stratified Analysis; p = 0.630, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.84 to 1.33]

5. Secondary Outcome: PFS as Determined by the Investigator Using RECIST v1.1 in the Tumor Cell (TC) 2/3 or Tumor-Infiltrating Immune Cell (IC) 2/3 Population
Description: PFS is defined as the time between the date of randomization and the date of first documented disease progression or death, whichever occurs first, in the Tumor Cell (TC) 2/3 or Tumor-Infiltrating Immune Cell (IC) 2/3 Population.
Time Frame: Up to approximately 30 months after first participant enrolled
Population: The PD-L1 TC2/3 or IC2/3 population is defined as particpants in the ITT population with PD-L1 TC2/3 or IC2/3 expression in baseline tumor tissue.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm C: Nab-Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 108 | 115 | 100
Months | 5.6 [5.1 to 5.7] | 8.4 [6.8 to 10.4] | 7.0 [5.6 to 8.3]
Statistical Analysis 1: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin; Test type: Superiority — Unstratified Analysis; p < .0001, Log Rank; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.40 to 0.72]
Statistical Analysis 2: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm A: Atezolizumab + Paclitaxel + Carboplatin; Test type: Superiority — Unstratified Analysis; p = 0.0018, Log Rank; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.45 to 0.84]

6. Secondary Outcome: PFS as Determined by the Investigator Using RECIST v1.1 in the TC1/2/3 or IC1/2/3 Population
Description: PFS is defined as the time between the date of randomization and the date of first documented disease progression or death, whichever occurs first, in the TC1/2/3 or IC1/2/3 Population.
Time Frame: Up to approximately 30 months after first participant enrolled
Population: The PD-L1 TC1/2/3 or IC1/2/3 population is defined as participants in the ITT population with PD-L1 TC1/2/3 or IC1/2/3 expression in baseline tumor tissue.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm C: Nab-Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 169 | 182 | 167
Months | 5.6 [5.3 to 5.7] | 7.1 [5.8 to 8.3] | 7.0 [5.6 to 8.3]
Statistical Analysis 1: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin; Test type: Superiority — Unstratified Analysis; p < .0001, Log Rank; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.48 to 0.77]
Statistical Analysis 2: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm A: Atezolizumab + Paclitaxel + Carboplatin; Test type: Superiority — Unstratified Analysis; p < .0001, Log Rank; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.48 to 0.77]

7. Secondary Outcome: OS in the TC2/3 or IC2/3 Population
Description: OS is defined as the time between the date of randomization and date of death from any cause, in the TC2/3 or IC2/3 Population.
Time Frame: Up to approximately 39 months after first participant enrolled
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm C: Nab-Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 108 | 115 | 100
Months | 14.5 [12.1 to 17.2] | 20.4 [13.8 to 24.1] | 14.8 [11.1 to 23.7]
Statistical Analysis 1: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm A: Atezolizumab + Paclitaxel + Carboplatin; Test type: Superiority — Unstratified Analysis; p = 0.0518, Log Rank; Hazard Ratio (HR) = 0.725, 95% CI 2-sided [0.524 to 1.004]
Statistical Analysis 2: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin; Test type: Superiority — Unstratified Analysis; p = 0.2841, Log Rank; Hazard Ratio (HR) = 0.832, 95% CI 2-sided [0.594 to 1.165]

8. Secondary Outcome: OS in the TC1/2/3 or IC1/2/3 Population
Description: OS is defined as the time between the date of randomization and date of death from any cause in the TC1/2/3 or IC1/2/3 Population.
Time Frame: Up to approximately 39 months after first participant enrolled
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm C: Nab-Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 169 | 182 | 167
Months | 15.0 [12.4 to 17.2] | 14.8 [12.1 to 19.6] | 14.9 [12.5 to 18.2]
Statistical Analysis 1: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm A: Atezolizumab + Paclitaxel + Carboplatin; Test type: Superiority — Unstratified Analysis; p = 0.2956, Log Rank; Hazard Ratio (HR) = 0.871, 95% CI 2-sided [0.671 to 1.129]
Statistical Analysis 2: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin; Test type: Superiority — Unstratified Analysis; p = 0.2473, Log Rank; Hazard Ratio (HR) = 0.861, 95% CI 2-sided [0.668 to 1.109]

9. Secondary Outcome: Percentage of Participants With Objective Response as Determined by the Investigator Using RECIST v1.1 in the ITT Population
Description: Proportion of participants with an objective response (CR or PR) in the ITT population.
Time Frame: Up to approximately 30 months after first participant enrolled
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Arm C: Nab-Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 339 | 342 | 337
Percentage of participants | 41.0 | 49.7 | 49.3
Statistical Analysis 1: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin; Test type: Superiority — Stratified Analysis; p = 0.0248, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.41, 95% CI 2-sided [1.04 to 1.91]
Statistical Analysis 2: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm A: Atezolizumab + Paclitaxel + Carboplatin; Test type: Superiority — Stratified Analysis; p = 0.0308, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.40, 95% CI 2-sided [1.03 to 1.90]

10. Secondary Outcome: Duration of Response as Determined by the Investigator Using RECIST v1.1 in the ITT Population
Description: Duration of response is defined as the time from the first documented objective response to documented PD or death from any cause, whichever occurred first, in the ITT Population.
Time Frame: Up to approximately 30 months after first participant enrolled
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm C: Nab-Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 139 | 170 | 166
Months | 5.2 [4.4 to 5.6] | 7.2 [6.8 to 9.5] | 7.0 [5.7 to 8.3]
Statistical Analysis 1: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin; Test type: Superiority — Unstratified Analysis; p < .0001, Log Rank; Hazard Ratio (HR) = 0.530, 95% CI 2-sided [0.408 to 0.689]
Statistical Analysis 2: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm A: Atezolizumab + Paclitaxel + Carboplatin; Test type: Superiority — Unstratified Analysis; p = 0.0007, Log Rank; Hazard Ratio (HR) = 0.640, 95% CI 2-sided [0.493 to 0.831]

11. Secondary Outcome: Event Free Rate at 1 and 2 Years in the ITT Population
Description: Event free rate at 1 and 2 years is defined as the proportion of participants alive at 1 and 2 years after randomization estimated using Kaplan-Meier (KM) methodology for the ITT population.
Time Frame: 1 and 2 years
Population: Participants still alive at 1 or 2 years after randomization from the ITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm C: Nab-Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 184 | 187 | 170
Percentage of participants
  1 Year | 56.28 | 56.34 | 52.30
  2 Year: number analyzed (Participants) | 49 | 68 | 50
  2 Year | 26.58 | 32.51 | 27.79
Statistical Analysis 1: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin; Event Free Rate (%) at Year 1; Test type: Superiority; p = 0.9871, Z-test; Difference in Event Free Rate = 0.06, 95% CI 2-sided [-7.48 to 7.61]
Statistical Analysis 2: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin; Event Free Rate (%) at Year 2; Test type: Superiority; p = 0.1133, Z-test; Difference in Event Free Rate = 5.93, 95% CI 2-sided [-1.41 to 13.26]
Statistical Analysis 3: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm A: Atezolizumab + Paclitaxel + Carboplatin; Event Free Rate (%) at Year 1; Test type: Superiority; p = 0.3072, Z-test; Difference in Event Free Rate = -3.97, 95% CI 2-sided [-11.60 to 3.65]
Statistical Analysis 4: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm A: Atezolizumab + Paclitaxel + Carboplatin; Event Free Rate (%) at Year 2; Test type: Superiority; p = 0.7430, Z-test; Difference in Event Free Rate = 1.21, 95% CI 2-sided [-6.01 to 8.42]

12. Secondary Outcome: Time to Deterioration (TTD) in Patient-reported Lung Cancer Symptoms Using EORTC QLQ-C30 Symptom Subscales in the ITT Population
Description: TTD in Patient-reported Lung Cancer Symptoms Using EORTC QLQ-C30 Symptom Subscales in the ITT Population. The EORTC QLQ-C30 is a validated and reliable self-report measure that consists of 30 questions that assess five aspects of patient functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, pain), global health/quality of life, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). EORTC scales and single-item measures will be linearly transformed so that each score has a range of 0-100. A high score for a functional scale represents a high or healthy level of functioning, and a high score for the global health status and HRQoL represents a high HRQoL; however, a high score for a symptom scale or item represents a high level of symptomatology or problems.
Time Frame: Up to approximately 30 months after first participant enrolled
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm C: Nab-Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 340 | 343 | 338
Months | 3.2 [2.6 to 4.1] | 4.2 [3.2 to 5.6] | 3.0 [2.6 to 3.9]
Statistical Analysis 1: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin; Test type: Superiority — Stratified Analysis; p = 0.0461, Log Rank; Hazard Ratio (HR) = 0.797, 95% CI 2-sided [0.638 to 0.996]
Statistical Analysis 2: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm A: Atezolizumab + Paclitaxel + Carboplatin; Test type: Superiority — Stratified Analysis; p = 0.7295, Log Rank; Hazard Ratio (HR) = 1.040, 95% CI 2-sided [0.834 to 1.296]

13. Secondary Outcome: TTD in Patient-reported Lung Cancer Symptoms Using EORTC QLQ-LC13 Symptom Subscales in the ITT Population
Description: TTD was documented for a 3-symptom composite endpoint using the following EORTC QLQ-LC13 symptom scores: cough, chest pain, and dyspnea multi--item scale. In this instance, symptom deterioration will be determined as a >= 10-point increase above baseline in any of the listed symptom scores, whichever occurs first (cough, chest pain, and dyspnea multi-item scale). Confirmed clinically meaningful symptom deterioration will need to be held for the original symptom; a >= 10-point increase above baseline in a symptom score must be held for at least two consecutive assessments or an initial>=10-point increase above baseline followed by death within 3 weeks from the last assessment. A >= 10-point change in the EORTC scale score is perceived by patients as clinically significant.
Time Frame: Up to approximately 30 months after the first participant enrolled
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm C: Nab-Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 340 | 343 | 338
Months | 2.6 [2.2 to 3.0] | 3.4 [2.7 to 5.1] | 2.8 [2.1 to 3.7]
Statistical Analysis 1: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin; Test type: Superiority — Stratified Analysis; p = 0.0942, Log Rank; Hazard Ratio (HR) = 0.828, 95% CI 2-sided [0.663 to 1.033]
Statistical Analysis 2: Comparison: Arm C: Nab-Paclitaxel + Carboplatin vs Arm A: Atezolizumab + Paclitaxel + Carboplatin; Test type: Superiority — Stratified Analysis; p = 0.7709, Log Rank; Hazard Ratio (HR) = 0.968, 95% CI 2-sided [0.776 to 1.207]

14. Secondary Outcome: Change From Baseline in Patient-reported Lung Cancer Symptoms Score Using the SILC Scale Symptom Severity Score in the ITT Population
Description: Change from baseline per SILC scale will be analyzed for each lung cancer symptoms scores. SILC questionnaire comprises 3 individual symptoms & are scored at individual symptom level, thus have a dyspnea score, chest pain score, & cough score. There are a total of 9 questions in SILC questionnaire, each question has a minimum value of 0 & maximum value of 4. Each individual symptom score is calculated as average of responses for symptom items. 'Chest pain' score is mean of question 1 & 2, 'Cough' score is mean of question 3 & 4 and 'Dyspnea' score is mean of question 5 to 9 in SILC questionnaire. An increase in score is suggestive of a worsening in symptomology. A score change of ≥0.3 points for dyspnea & cough symptom scores is considered to be clinically significant; whereas a score change of ≥0.5 points for chest pain score is considered to be clinically significant. (Note: PD=progression of disease)
Time Frame: Baseline up to approximately 30 months after first participant enrolled
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm C: Nab-Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 189 | 215 | 195
Units on a scale
  Chest Pain, Week 1: number analyzed (Participants) | 171 | 192 | 166
  Chest Pain, Week 1 | 0.04 (0.93) | 0.14 (0.87) | 0.44 (1.03)
  Chest Pain, Week 2: number analyzed (Participants) | 160 | 186 | 165
  Chest Pain, Week 2 | -0.08 (0.89) | 0.09 (0.98) | 0.28 (1.00)
  Chest Pain, Week 3: number analyzed (Participants) | 165 | 175 | 165
  Chest Pain, Week 3 | -0.14 (0.95) | -0.03 (0.78) | -0.05 (1.00)
  Chest Pain, Week 4: number analyzed (Participants) | 157 | 173 | 169
  Chest Pain, Week 4 | -0.19 (0.98) | -0.05 (0.98) | 0.09 (1.12)
  Chest Pain, Week 5: number analyzed (Participants) | 160 | 172 | 159
  Chest Pain, Week 5 | -0.17 (1.10) | -0.08 (0.99) | -0.16 (1.09)
  Chest Pain, Week 6: number analyzed (Participants) | 151 | 170 | 161
  Chest Pain, Week 6 | -0.35 (1.08) | -0.13 (0.99) | -0.20 (1.02)
  Chest Pain, Week 7: number analyzed (Participants) | 138 | 166 | 143
  Chest Pain, Week 7 | -0.38 (1.12) | -0.18 (0.92) | -0.14 (1.16)
  Chest Pain, Week 8: number analyzed (Participants) | 140 | 162 | 152
  Chest Pain, Week 8 | -0.35 (1.12) | -0.17 (1.02) | -0.17 (1.09)
  Chest Pain, Week 9: number analyzed (Participants) | 135 | 162 | 143
  Chest Pain, Week 9 | -0.36 (1.00) | -0.19 (0.97) | -0.21 (1.10)
  Chest Pain, Week 10: number analyzed (Participants) | 133 | 158 | 146
  Chest Pain, Week 10 | -0.20 (1.09) | -0.16 (1.00) | -0.08 (1.19)
  Chest Pain, Week 11: number analyzed (Participants) | 132 | 157 | 137
  Chest Pain, Week 11 | -0.27 (1.08) | -0.24 (0.91) | -0.09 (1.16)
  Chest Pain, Week 12: number analyzed (Participants) | 128 | 151 | 136
  Chest Pain, Week 12 | -0.34 (1.05) | -0.21 (1.01) | -0.30 (1.05)
  Chest Pain, Week 13: number analyzed (Participants) | 117 | 144 | 130
  Chest Pain, Week 13 | -0.31 (1.24) | -0.22 (1.02) | -0.17 (1.10)
  Chest Pain, Week 14: number analyzed (Participants) | 105 | 139 | 138
  Chest Pain, Week 14 | -0.32 (1.18) | -0.24 (0.88) | -0.15 (1.13)
  Chest Pain, Week 15: number analyzed (Participants) | 97 | 143 | 132
  Chest Pain, Week 15 | -0.45 (1.19) | -0.28 (0.99) | -0.17 (1.00)
  Chest Pain, Week 16: number analyzed (Participants) | 102 | 138 | 121
  Chest Pain, Week 16 | -0.28 (1.10) | -0.14 (1.00) | -0.23 (1.10)
  Chest Pain, Week 17: number analyzed (Participants) | 101 | 135 | 129
  Chest Pain, Week 17 | -0.32 (1.11) | -0.17 (0.99) | -0.24 (1.10)
  Chest Pain, Week 18: number analyzed (Participants) | 93 | 141 | 129
  Chest Pain, Week 18 | -0.28 (1.08) | -0.13 (0.99) | -0.17 (1.09)
  Chest Pain, Week 19: number analyzed (Participants) | 85 | 129 | 118
  Chest Pain, Week 19 | -0.18 (1.09) | -0.10 (0.99) | -0.16 (1.07)
  Chest Pain, Week 20: number analyzed (Participants) | 75 | 130 | 114
  Chest Pain, Week 20 | -0.23 (1.07) | -0.15 (0.94) | -0.17 (1.13)
  Chest Pain, Week 21: number analyzed (Participants) | 69 | 129 | 113
  Chest Pain, Week 21 | -0.37 (1.02) | -0.07 (1.02) | -0.18 (1.14)
  Chest Pain, Week 22: number analyzed (Participants) | 79 | 125 | 109
  Chest Pain, Week 22 | -0.27 (1.18) | -0.08 (1.01) | -0.14 (1.16)
  Chest Pain, Week 23: number analyzed (Participants) | 70 | 128 | 106
  Chest Pain, Week 23 | -0.29 (1.16) | 0.04 (0.96) | -0.10 (1.07)
  Chest Pain, Week 24: number analyzed (Participants) | 67 | 121 | 105
  Chest Pain, Week 24 | -0.43 (1.15) | -0.15 (0.97) | -0.17 (1.14)
  Chest Pain, Week 25: number analyzed (Participants) | 48 | 118 | 104
  Chest Pain, Week 25 | -0.25 (1.24) | -0.17 (1.06) | -0.20 (1.10)
  Chest Pain, Week 26: number analyzed (Participants) | 48 | 111 | 99
  Chest Pain, Week 26 | -0.50 (1.20) | -0.06 (1.08) | -0.11 (1.09)
  Chest Pain, Week 27: number analyzed (Participants) | 42 | 110 | 95
  Chest Pain, Week 27 | -0.35 (1.29) | -0.17 (1.03) | 0.04 (1.14)
  Chest Pain, Week 28: number analyzed (Participants) | 41 | 103 | 88
  Chest Pain, Week 28 | -0.22 (1.27) | -0.12 (1.09) | -0.19 (1.24)
  Chest Pain, Week 29: number analyzed (Participants) | 38 | 100 | 89
  Chest Pain, Week 29 | -0.30 (1.23) | -0.11 (0.96) | -0.18 (1.11)
  Chest Pain, Week 30: number analyzed (Participants) | 46 | 104 | 86
  Chest Pain, Week 30 | -0.15 (1.36) | -0.21 (1.02) | -0.08 (1.09)
  Chest Pain, Week 31: number analyzed (Participants) | 35 | 97 | 77
  Chest Pain, Week 31 | -0.49 (1.25) | -0.16 (0.99) | -0.15 (1.08)
  Chest Pain, Week 32: number analyzed (Participants) | 29 | 91 | 70
  Chest Pain, Week 32 | -0.29 (1.16) | -0.15 (0.88) | -0.16 (1.01)
  Chest Pain, Week 33: number analyzed (Participants) | 29 | 93 | 68
  Chest Pain, Week 33 | -0.29 (1.35) | -0.20 (0.97) | -0.10 (1.09)
  Chest Pain, Week 34: number analyzed (Participants) | 33 | 92 | 73
  Chest Pain, Week 34 | -0.15 (1.42) | -0.04 (0.89) | 0.02 (1.16)
  Chest Pain, Week 35: number analyzed (Participants) | 33 | 90 | 72
  Chest Pain, Week 35 | -0.26 (1.31) | -0.14 (0.88) | -0.19 (1.09)
  Chest Pain, Week 36: number analyzed (Participants) | 31 | 83 | 64
  Chest Pain, Week 36 | -0.24 (1.34) | -0.06 (0.88) | -0.06 (1.12)
  Chest Pain, Week 37: number analyzed (Participants) | 24 | 84 | 65
  Chest Pain, Week 37 | -0.27 (1.37) | 0.05 (1.06) | -0.08 (1.08)
  Chest Pain, Week 38: number analyzed (Participants) | 24 | 86 | 65
  Chest Pain, Week 38 | -0.19 (1.30) | -0.09 (0.97) | -0.14 (1.13)
  Chest Pain, Week 39: number analyzed (Participants) | 25 | 75 | 68
  Chest Pain, Week 39 | -0.06 (1.53) | -0.18 (0.96) | -0.13 (1.13)
  Chest Pain, Week 40: number analyzed (Participants) | 24 | 74 | 62
  Chest Pain, Week 40 | 0.06 (1.31) | -0.11 (0.85) | -0.06 (1.01)
  Chest Pain, Week 41: number analyzed (Participants) | 22 | 69 | 60
  Chest Pain, Week 41 | 0.14 (1.21) | -0.14 (0.92) | -0.13 (1.05)
  Chest Pain, Week 42: number analyzed (Participants) | 24 | 77 | 60
  Chest Pain, Week 42 | -0.10 (1.50) | -0.05 (0.94) | -0.11 (1.02)
  Chest Pain, Week 43: number analyzed (Participants) | 23 | 72 | 58
  Chest Pain, Week 43 | 0.13 (1.59) | -0.08 (0.99) | 0.05 (1.13)
  Chest Pain, Week 44: number analyzed (Participants) | 20 | 93 | 60
  Chest Pain, Week 44 | -0.08 (1.52) | -0.25 (0.99) | -0.10 (1.07)
  Chest Pain, Week 45: number analyzed (Participants) | 20 | 64 | 51
  Chest Pain, Week 45 | 0.15 (1.70) | -0.21 (0.97) | -0.05 (1.20)
  Chest Pain, Week 46: number analyzed (Participants) | 20 | 61 | 53
  Chest Pain, Week 46 | 0.00 (1.39) | -0.16 (1.04) | -0.07 (1.33)
  Chest Pain, Week 47: number analyzed (Participants) | 20 | 64 | 48
  Chest Pain, Week 47 | 0.18 (1.29) | -0.16 (0.99) | 0.04 (1.29)
  Chest Pain, Week 48: number analyzed (Participants) | 19 | 62 | 52
  Chest Pain, Week 48 | -0.08 (1.53) | -0.17 (0.97) | 0.00 (1.32)
  Chest Pain, Week 49: number analyzed (Participants) | 13 | 57 | 45
  Chest Pain, Week 49 | -0.23 (1.59) | -0.24 (1.05) | -0.09 (1.31)
  Chest Pain, Week 50: number analyzed (Participants) | 15 | 60 | 45
  Chest Pain, Week 50 | 0.00 (1.73) | -0.17 (0.98) | -0.14 (1.36)
  Chest Pain, Week 51: number analyzed (Participants) | 11 | 58 | 37
  Chest Pain, Week 51 | 0.55 (1.39) | -0.16 (1.07) | -0.19 (1.24)
  Chest Pain, Week 52: number analyzed (Participants) | 13 | 58 | 43
  Chest Pain, Week 52 | 0.15 (1.30) | -0.09 (0.98) | 0.02 (1.30)
  Chest Pain, Week 53: number analyzed (Participants) | 14 | 53 | 35
  Chest Pain, Week 53 | 0.18 (1.27) | -0.12 (0.95) | -0.20 (1.22)
  Chest Pain, Week 54: number analyzed (Participants) | 13 | 56 | 36
  Chest Pain, Week 54 | 0.08 (1.17) | -0.18 (0.92) | -0.24 (1.34)
  Chest Pain, Week 55: number analyzed (Participants) | 12 | 47 | 36
  Chest Pain, Week 55 | 0.21 (1.37) | -0.11 (0.79) | -0.15 (1.19)
  Chest Pain, Week 56: number analyzed (Participants) | 11 | 50 | 36
  Chest Pain, Week 56 | 0.05 (1.39) | -0.22 (0.91) | -0.08 (1.36)
  Chest Pain, Week 57: number analyzed (Participants) | 10 | 52 | 33
  Chest Pain, Week 57 | 0.05 (1.46) | -0.22 (0.95) | -0.27 (1.22)
  Chest Pain, Week 58: number analyzed (Participants) | 8 | 45 | 29
  Chest Pain, Week 58 | 0.13 (1.25) | -0.22 (0.86) | -0.24 (1.12)
  Chest Pain, Week 59: number analyzed (Participants) | 11 | 47 | 27
  Chest Pain, Week 59 | 0.00 (1.32) | -0.20 (1.01) | -0.28 (1.17)
  Chest Pain, Week 60: number analyzed (Participants) | 11 | 41 | 31
  Chest Pain, Week 60 | 0.09 (1.59) | -0.27 (0.97) | -0.26 (1.22)
  Chest Pain, Week 61: number analyzed (Participants) | 9 | 40 | 28
  Chest Pain, Week 61 | 0.61 (1.29) | -0.23 (0.83) | -0.34 (1.23)
  Chest Pain, Week 62: number analyzed (Participants) | 10 | 39 | 25
  Chest Pain, Week 62 | 0.05 (1.34) | -0.03 (1.00) | -0.36 (0.96)
  Chest Pain, Week 63: number analyzed (Participants) | 8 | 42 | 22
  Chest Pain, Week 63 | -0.44 (1.21) | -0.12 (0.92) | -0.55 (1.13)
  Chest Pain, Week 64: number analyzed (Participants) | 8 | 42 | 18
  Chest Pain, Week 64 | 0.19 (1.49) | -0.13 (0.99) | -0.42 (1.33)
  Chest Pain, Week 65: number analyzed (Participants) | 6 | 39 | 20
  Chest Pain, Week 65 | 0.25 (1.37) | -0.13 (0.95) | -0.25 (1.21)
  Chest Pain, Week 66: number analyzed (Participants) | 6 | 37 | 19
  Chest Pain, Week 66 | 0.42 (1.53) | 0.00 (1.26) | -0.47 (1.18)
  Chest Pain, Week 67: number analyzed (Participants) | 5 | 33 | 20
  Chest Pain, Week 67 | -0.50 (1.27) | -0.08 (1.04) | -0.43 (1.27)
  Chest Pain, Week 68: number analyzed (Participants) | 6 | 33 | 19
  Chest Pain, Week 68 | 0.08 (1.77) | -0.09 (1.02) | -0.53 (1.23)
  Chest Pain, Week 69: number analyzed (Participants) | 5 | 31 | 18
  Chest Pain, Week 69 | 0.70 (1.60) | -0.15 (1.08) | -0.03 (1.14)
  Chest Pain, Week 70: number analyzed (Participants) | 5 | 32 | 19
  Chest Pain, Week 70 | 0.30 (1.79) | -0.06 (0.97) | -0.32 (1.08)
  Chest Pain, Week 71: number analyzed (Participants) | 6 | 27 | 15
  Chest Pain, Week 71 | 0.08 (1.72) | -0.13 (0.91) | -0.43 (1.22)
  Chest Pain, Week 72: number analyzed (Participants) | 6 | 27 | 18
  Chest Pain, Week 72 | 0.25 (1.70) | -0.20 (0.94) | -0.14 (1.00)
  Chest Pain, Week 73: number analyzed (Participants) | 6 | 27 | 13
  Chest Pain, Week 73 | 0.42 (1.53) | -0.02 (1.09) | -0.08 (1.27)
  Chest Pain, Week 74: number analyzed (Participants) | 7 | 29 | 12
  Chest Pain, Week 74 | 0.43 (1.62) | -0.10 (1.14) | -0.38 (1.21)
  Chest Pain, Week 75: number analyzed (Participants) | 6 | 24 | 12
  Chest Pain, Week 75 | 0.25 (1.70) | -0.17 (0.89) | -0.21 (1.18)
  Chest Pain, Week 76: number analyzed (Participants) | 6 | 23 | 14
  Chest Pain, Week 76 | 0.00 (1.76) | -0.02 (1.03) | -0.21 (1.25)
  Chest Pain, Week 77: number analyzed (Participants) | 6 | 22 | 10
  Chest Pain, Week 77 | 0.00 (1.76) | 0.00 (1.15) | -0.05 (1.21)
  Chest Pain, Week 78: number analyzed (Participants) | 7 | 22 | 11
  Chest Pain, Week 78 | 0.07 (1.62) | -0.11 (1.11) | 0.00 (1.02)
  Chest Pain, Week 79: number analyzed (Participants) | 6 | 24 | 9
  Chest Pain, Week 79 | 0.08 (1.72) | -0.13 (0.86) | 0.17 (0.94)
  Chest Pain, Week 80: number analyzed (Participants) | 7 | 20 | 11
  Chest Pain, Week 80 | 0.14 (1.65) | -0.35 (0.99) | 0.09 (1.14)
  Chest Pain, Week 81: number analyzed (Participants) | 6 | 18 | 9
  Chest Pain, Week 81 | 0.25 (1.70) | -0.25 (0.90) | 0.22 (0.97)
  Chest Pain, Week 82: number analyzed (Participants) | 7 | 21 | 9
  Chest Pain, Week 82 | 0.07 (1.62) | -0.31 (1.03) | 0.22 (1.12)
  Chest Pain, Week 83: number analyzed (Participants) | 5 | 19 | 10
  Chest Pain, Week 83 | 0.00 (1.77) | -0.32 (1.03) | -0.05 (1.01)
  Chest Pain, Week 84: number analyzed (Participants) | 5 | 15 | 10
  Chest Pain, Week 84 | 0.00 (1.84) | -0.33 (1.08) | 0.35 (1.00)
  Chest Pain, Week 85: number analyzed (Participants) | 4 | 17 | 10
  Chest Pain, Week 85 | 1.13 (1.31) | -0.35 (1.03) | 0.30 (1.14)
  Chest Pain, Week 86: number analyzed (Participants) | 3 | 15 | 6
  Chest Pain, Week 86 | 1.33 (1.53) | -0.37 (0.95) | 0.33 (1.37)
  Chest Pain, Week 87: number analyzed (Participants) | 3 | 12 | 8
  Chest Pain, Week 87 | 1.00 (1.73) | -0.25 (1.10) | 0.13 (0.99)
  Chest Pain, Week 88: number analyzed (Participants) | 3 | 15 | 7
  Chest Pain, Week 88 | 0.83 (1.44) | -0.20 (1.22) | 0.00 (1.00)
  Chest Pain, Week 89: number analyzed (Participants) | 3 | 14 | 7
  Chest Pain, Week 89 | 0.67 (2.08) | -0.14 (1.08) | -0.29 (1.25)
  Chest Pain, Week 90: number analyzed (Participants) | 3 | 13 | 7
  Chest Pain, Week 90 | 0.67 (2.08) | -0.04 (1.25) | 0.00 (1.29)
  Chest Pain, Week 91: number analyzed (Participants) | 3 | 13 | 7
  Chest Pain, Week 91 | 1.17 (1.61) | -0.42 (1.13) | 0.14 (1.07)
  Chest Pain, Week 92: number analyzed (Participants) | 4 | 13 | 8
  Chest Pain, Week 92 | 0.88 (1.44) | -0.15 (1.20) | 0.19 (1.25)
  Chest Pain, Week 93: number analyzed (Participants) | 2 | 13 | 10
  Chest Pain, Week 93 | 1.50 (2.12) | 0.00 (1.24) | -0.05 (1.01)
  Chest Pain, Week 94: number analyzed (Participants) | 3 | 11 | 8
  Chest Pain, Week 94 | 0.67 (2.08) | -0.23 (1.35) | 0.00 (1.20)
  Chest Pain, Week 95: number analyzed (Participants) | 3 | 11 | 8
  Chest Pain, Week 95 | 0.67 (2.08) | 0.14 (1.19) | 0.25 (1.00)
  Chest Pain, Week 96: number analyzed (Participants) | 3 | 11 | 8
  Chest Pain, Week 96 | 1.17 (1.61) | 0.09 (1.53) | 0.19 (0.92)
  Chest Pain, Week 97: number analyzed (Participants) | 3 | 11 | 9
  Chest Pain, Week 97 | 1.17 (1.61) | -0.18 (1.54) | -0.11 (1.17)
  Chest Pain, Week 98: number analyzed (Participants) | 3 | 10 | 7
  Chest Pain, Week 98 | 0.83 (2.02) | 0.05 (1.48) | 0.00 (1.00)
  Chest Pain, Week 99: number analyzed (Participants) | 3 | 10 | 7
  Chest Pain, Week 99 | 0.67 (2.08) | 0.00 (1.53) | 0.07 (1.02)
  Chest Pain, Week 100: number analyzed (Participants) | 2 | 10 | 8
  Chest Pain, Week 100 | 1.25 (1.77) | -0.15 (1.43) | 0.00 (1.20)
  Chest Pain, Week 101: number analyzed (Participants) | 3 | 10 | 7
  Chest Pain, Week 101 | 1.17 (1.61) | -0.10 (1.54) | 0.21 (0.99)
  Chest Pain, Week 102: number analyzed (Participants) | 3 | 6 | 6
  Chest Pain, Week 102 | 1.00 (1.32) | -0.25 (0.88) | 0.08 (1.11)
  Chest Pain, Week 103: number analyzed (Participants) | 2 | 9 | 6
  Chest Pain, Week 103 | -0.50 (0.71) | -0.56 (1.04) | 0.17 (1.17)
  Chest Pain, Week 104: number analyzed (Participants) | 2 | 8 | 4
  Chest Pain, Week 104 | 0.25 (0.35) | -0.56 (1.05) | 0.00 (1.41)
  Chest Pain, Week 105: number analyzed (Participants) | 2 | 6 | 6
  Chest Pain, Week 105 | 0.50 (0.00) | -0.50 (0.84) | 0.00 (1.10)
  Chest Pain, Week 106: number analyzed (Participants) | 2 | 9 | 5
  Chest Pain, Week 106 | 0.00 (0.00) | -0.72 (1.06) | -0.40 (1.14)
  Chest Pain, Week 107: number analyzed (Participants) | 2 | 7 | 4
  Chest Pain, Week 107 | 0.25 (0.35) | -0.57 (1.17) | -0.50 (0.58)
  Chest Pain, Week 108: number analyzed (Participants) | 2 | 5 | 4
  Chest Pain, Week 108 | 0.25 (0.35) | -0.30 (1.25) | -0.38 (0.75)
  Chest Pain, Week 109: number analyzed (Participants) | 2 | 5 | 2
  Chest Pain, Week 109 | -0.50 (0.71) | -0.90 (1.24) | 0.25 (1.77)
  Chest Pain, Week 110: number analyzed (Participants) | 2 | 3 | 4
  Chest Pain, Week 110 | 0.00 (0.71) | -0.50 (1.32) | -0.38 (1.11)
  Chest Pain, Week 111: number analyzed (Participants) | 2 | 4 | 4
  Chest Pain, Week 111 | 0.25 (0.35) | -0.25 (1.26) | -0.38 (0.48)
  Chest Pain, Week 112: number analyzed (Participants) | 2 | 3 | 2
  Chest Pain, Week 112 | 0.50 (0.00) | -0.67 (1.15) | -1.00 (0.00)
  Chest Pain, Week 113: number analyzed (Participants) | 1 | 4 | 3
  Chest Pain, Week 113 | 0.00 | -0.50 (1.00) | -0.67 (0.58)
  Chest Pain, Week 114: number analyzed (Participants) | 2 | 3 | 2
  Chest Pain, Week 114 | -0.25 (1.06) | -0.50 (1.32) | -1.00 (0.00)
  Chest Pain, Week 115: number analyzed (Participants) | 2 | 4 | 3
  Chest Pain, Week 115 | -0.25 (1.06) | -0.50 (1.00) | -0.67 (0.58)
  Chest Pain, Week 116: number analyzed (Participants) | 2 | 3 | 3
  Chest Pain, Week 116 | -0.50 (0.71) | -0.67 (1.15) | -0.67 (0.58)
  Chest Pain, Week 117: number analyzed (Participants) | 2 | 2 | 2
  Chest Pain, Week 117 | -0.25 (1.06) | -1.00 (1.41) | -1.00 (0.00)
  Chest Pain, Week 118: number analyzed (Participants) | 1 | 1 | 2
  Chest Pain, Week 118 | 0.00 | 0.00 | -1.00 (0.00)
  Chest Pain, Week 119: number analyzed (Participants) | 0 | 1 | 2
  Chest Pain, Week 119 |  | 0.00 | -1.00 (0.00)
  Chest Pain, Week 120: number analyzed (Participants) | 0 | 1 | 2
  Chest Pain, Week 120 |  | 0.00 | -1.00 (0.00)
  Chest Pain, Week 121: number analyzed (Participants) | 0 | 1 | 2
  Chest Pain, Week 121 |  | 0.00 | -1.00 (0.00)
  Chest Pain, Week 122: number analyzed (Participants) | 0 | 1 | 2
  Chest Pain, Week 122 |  | 0.00 | -1.00 (0.00)
  Chest Pain, Week 123: number analyzed (Participants) | 0 | 1 | 1
  Chest Pain, Week 123 |  | 0.00 | -1.00
  Chest Pain, Week 124: number analyzed (Participants) | 0 | 1 | 1
  Chest Pain, Week 124 |  | 0.00 | -0.50
  Chest Pain, Week 125: number analyzed (Participants) | 0 | 0 | 1
  Chest Pain, Week 125 |  |  | -0.50
  Chest Pain, Week 126: number analyzed (Participants) | 0 | 0 | 1
  Chest Pain, Week 126 |  |  | -0.50
  Chest Pain, Week 127: number analyzed (Participants) | 0 | 0 | 1
  Chest Pain, Week 127 |  |  | -1.00
  Chest Pain, Time of First Pd: number analyzed (Participants) | 103 | 107 | 106
  Chest Pain, Time of First Pd | -0.19 (1.13) | 0.10 (1.12) | -0.11 (1.21)
  Chest Pain, Time of Last Tx Dose: number analyzed (Participants) | 161 | 172 | 151
  Chest Pain, Time of Last Tx Dose | -0.18 (1.06) | 0.01 (1.09) | 0.05 (1.14)
  Chest Pain, Survival Follow-Up Month 1: number analyzed (Participants) | 86 | 0 | 0
  Chest Pain, Survival Follow-Up Month 1 | 0.03 (1.30) |  |
  Chest Pain, Survival Follow-Up Month 2: number analyzed (Participants) | 52 | 0 | 0
  Chest Pain, Survival Follow-Up Month 2 | -0.10 (1.23) |  |
  Chest Pain, Survival Follow-Up Month 3: number analyzed (Participants) | 40 | 0 | 0
  Chest Pain, Survival Follow-Up Month 3 | -0.09 (1.13) |  |
  Chest Pain, Survival Follow-Up Month 4: number analyzed (Participants) | 32 | 0 | 0
  Chest Pain, Survival Follow-Up Month 4 | -0.13 (1.15) |  |
  Chest Pain, Survival Follow-Up Month 5: number analyzed (Participants) | 26 | 0 | 0
  Chest Pain, Survival Follow-Up Month 5 | -0.02 (1.34) |  |
  Chest Pain, Survival Follow-Up Month 6: number analyzed (Participants) | 23 | 0 | 0
  Chest Pain, Survival Follow-Up Month 6 | -0.22 (0.99) |  |
  Chest Pain, Survival Follow-Up Month 7: number analyzed (Participants) | 3 | 0 | 0
  Chest Pain, Survival Follow-Up Month 7 | 0.33 (0.58) |  |
  Chest Pain, Survival Follow-Up Month 8: number analyzed (Participants) | 2 | 0 | 0
  Chest Pain, Survival Follow-Up Month 8 | -0.75 (1.06) |  |
  Cough, Week 1: number analyzed (Participants) | 171 | 192 | 166
  Cough, Week 1 | 0.01 (0.78) | 0.03 (0.82) | -0.02 (0.74)
  Cough, Week 2: number analyzed (Participants) | 160 | 186 | 165
  Cough, Week 2 | -0.02 (0.91) | 0.00 (0.90) | 0.17 (0.87)
  Cough, Week 3: number analyzed (Participants) | 165 | 175 | 165
  Cough, Week 3 | -0.09 (0.90) | -0.10 (1.03) | -0.08 (0.95)
  Cough, Week 4: number analyzed (Participants) | 157 | 173 | 169
  Cough, Week 4 | -0.26 (0.92) | -0.16 (1.04) | -0.33 (1.07)
  Cough, Week 5: number analyzed (Participants) | 160 | 172 | 159
  Cough, Week 5 | -0.18 (1.02) | -0.24 (1.08) | -0.19 (1.13)
  Cough, Week 6: number analyzed (Participants) | 151 | 170 | 161
  Cough, Week 6 | -0.27 (1.05) | -0.22 (1.01) | -0.35 (1.11)
  Cough, Week 7: number analyzed (Participants) | 138 | 166 | 143
  Cough, Week 7 | -0.27 (1.06) | -0.27 (1.07) | -0.47 (1.11)
  Cough, Week 8: number analyzed (Participants) | 140 | 162 | 152
  Cough, Week 8 | -0.26 (1.11) | -0.26 (0.97) | -0.36 (1.09)
  Cough, Week 9: number analyzed (Participants) | 135 | 162 | 143
  Cough, Week 9 | -0.32 (1.16) | -0.27 (1.01) | -0.34 (1.09)
  Cough, Week 10: number analyzed (Participants) | 133 | 158 | 146
  Cough, Week 10 | -0.28 (1.02) | -0.28 (1.09) | -0.42 (1.08)
  Cough, Week 11: number analyzed (Participants) | 132 | 157 | 137
  Cough, Week 11 | -0.31 (0.98) | -0.27 (1.14) | -0.50 (1.06)
  Cough, Week 12: number analyzed (Participants) | 128 | 151 | 136
  Cough, Week 12 | -0.30 (1.08) | -0.25 (1.13) | -0.46 (1.06)
  Cough, Week 13: number analyzed (Participants) | 117 | 144 | 130
  Cough, Week 13 | -0.23 (1.14) | -0.28 (1.17) | -0.46 (1.10)
  Cough, Week 14: number analyzed (Participants) | 105 | 139 | 138
  Cough, Week 14 | -0.31 (1.09) | -0.29 (1.13) | -0.50 (1.16)
  Cough, Week 15: number analyzed (Participants) | 97 | 143 | 132
  Cough, Week 15 | -0.39 (1.11) | -0.23 (1.03) | -0.47 (1.18)
  Cough, Week 16: number analyzed (Participants) | 102 | 138 | 121
  Cough, Week 16 | -0.19 (1.19) | -0.18 (1.14) | -0.52 (1.25)
  Cough, Week 17: number analyzed (Participants) | 101 | 135 | 129
  Cough, Week 17 | -0.18 (1.08) | -0.21 (1.06) | -0.48 (1.16)
  Cough, Week 18: number analyzed (Participants) | 93 | 141 | 129
  Cough, Week 18 | -0.26 (1.09) | -0.34 (1.12) | -0.48 (1.05)
  Cough, Week 19: number analyzed (Participants) | 85 | 129 | 118
  Cough, Week 19 | -0.29 (1.05) | -0.29 (1.12) | -0.37 (1.04)
  Cough, Week 20: number analyzed (Participants) | 75 | 130 | 114
  Cough, Week 20 | -0.29 (1.09) | -0.24 (1.00) | -0.51 (1.15)
  Cough, Week 21: number analyzed (Participants) | 69 | 129 | 113
  Cough, Week 21 | -0.36 (1.01) | -0.26 (1.06) | -0.46 (1.09)
  Cough, Week 22: number analyzed (Participants) | 79 | 125 | 109
  Cough, Week 22 | -0.25 (1.13) | -0.27 (1.09) | -0.44 (1.11)
  Cough, Week 23: number analyzed (Participants) | 70 | 128 | 106
  Cough, Week 23 | -0.26 (1.19) | -0.30 (1.07) | -0.45 (1.17)
  Cough, Week 24: number analyzed (Participants) | 67 | 121 | 105
  Cough, Week 24 | -0.28 (1.14) | -0.33 (1.00) | -0.46 (1.11)
  Cough, Week 25: number analyzed (Participants) | 48 | 118 | 104
  Cough, Week 25 | -0.28 (1.18) | -0.31 (1.09) | -0.52 (1.06)
  Cough, Week 26: number analyzed (Participants) | 48 | 111 | 99
  Cough, Week 26 | -0.41 (1.08) | -0.32 (1.09) | -0.54 (1.24)
  Cough, Week 27: number analyzed (Participants) | 42 | 110 | 95
  Cough, Week 27 | -0.27 (1.11) | -0.39 (1.10) | -0.31 (1.20)
  Cough, Week 28: number analyzed (Participants) | 41 | 103 | 88
  Cough, Week 28 | -0.34 (1.10) | -0.36 (1.07) | -0.52 (1.21)
  Cough, Week 29: number analyzed (Participants) | 38 | 100 | 89
  Cough, Week 29 | -0.38 (1.15) | -0.33 (1.06) | -0.48 (1.13)
  Cough, Week 30: number analyzed (Participants) | 46 | 104 | 86
  Cough, Week 30 | -0.29 (1.15) | -0.31 (1.02) | -0.54 (1.14)
  Cough, Week 31: number analyzed (Participants) | 35 | 97 | 77
  Cough, Week 31 | -0.46 (1.14) | -0.34 (1.11) | -0.49 (1.10)
  Cough, Week 32: number analyzed (Participants) | 29 | 91 | 70
  Cough, Week 32 | -0.17 (0.98) | -0.41 (1.02) | -0.53 (1.04)
  Cough, Week 33: number analyzed (Participants) | 29 | 93 | 68
  Cough, Week 33 | -0.31 (1.11) | -0.35 (0.97) | -0.53 (1.13)
  Cough, Week 34: number analyzed (Participants) | 33 | 92 | 73
  Cough, Week 34 | -0.03 (0.93) | -0.34 (0.84) | -0.41 (1.14)
  Cough, Week 35: number analyzed (Participants) | 33 | 90 | 72
  Cough, Week 35 | -0.14 (1.01) | -0.38 (0.91) | -0.47 (1.05)
  Cough, Week 36: number analyzed (Participants) | 31 | 83 | 64
  Cough, Week 36 | -0.05 (0.93) | -0.39 (0.96) | -0.43 (0.99)
  Cough, Week 37: number analyzed (Participants) | 24 | 84 | 65
  Cough, Week 37 | -0.08 (1.11) | -0.22 (0.94) | -0.54 (1.12)
  Cough, Week 38: number analyzed (Participants) | 24 | 86 | 65
  Cough, Week 38 | 0.02 (1.09) | -0.36 (0.97) | -0.45 (1.16)
  Cough, Week 39: number analyzed (Participants) | 25 | 75 | 68
  Cough, Week 39 | 0.00 (1.05) | -0.46 (1.05) | -0.50 (1.06)
  Cough, Week 40: number analyzed (Participants) | 24 | 74 | 62
  Cough, Week 40 | 0.10 (1.12) | -0.39 (1.04) | -0.47 (1.02)
  Cough, Week 41: number analyzed (Participants) | 22 | 69 | 60
  Cough, Week 41 | 0.07 (1.21) | -0.43 (1.10) | -0.58 (1.06)
  Cough, Week 42: number analyzed (Participants) | 24 | 77 | 60
  Cough, Week 42 | -0.04 (1.16) | -0.41 (1.05) | -0.68 (1.05)
  Cough, Week 43: number analyzed (Participants) | 23 | 72 | 58
  Cough, Week 43 | -0.02 (0.87) | -0.38 (1.04) | -0.45 (0.99)
  Cough, Week 44: number analyzed (Participants) | 20 | 63 | 60
  Cough, Week 44 | -0.05 (1.24) | -0.48 (1.21) | -0.56 (1.09)
  Cough, Week 45: number analyzed (Participants) | 20 | 64 | 51
  Cough, Week 45 | 0.10 (1.24) | -0.32 (1.11) | -0.69 (1.00)
  Cough, Week 46: number analyzed (Participants) | 20 | 61 | 53
  Cough, Week 46 | 0.03 (0.95) | -0.38 (1.11) | -0.67 (1.10)
  Cough, Week 47: number analyzed (Participants) | 20 | 64 | 48
  Cough, Week 47 | 0.10 (1.15) | -0.38 (1.13) | -0.54 (0.97)
  Cough, Week 48: number analyzed (Participants) | 19 | 62 | 52
  Cough, Week 48 | 0.00 (1.22) | -0.41 (1.09) | -0.55 (1.09)
  Cough, Week 49: number analyzed (Participants) | 13 | 57 | 45
  Cough, Week 49 | -0.12 (1.04) | -0.44 (1.10) | -0.63 (1.06)
  Cough, Week 50: number analyzed (Participants) | 15 | 60 | 45
  Cough, Week 50 | 0.23 (0.98) | -0.29 (1.16) | -0.72 (1.07)
  Cough, Week 51: number analyzed (Participants) | 11 | 58 | 37
  Cough, Week 51 | 0.05 (0.88) | -0.22 (1.20) | -0.69 (1.11)
  Cough, Week 52: number analyzed (Participants) | 13 | 58 | 43
  Cough, Week 52 | 0.12 (0.79) | -0.33 (1.19) | -0.64 (1.03)
  Cough, Week 53: number analyzed (Participants) | 14 | 53 | 35
  Cough, Week 53 | 0.21 (0.78) | -0.28 (1.14) | -0.53 (1.19)
  Cough, Week 54: number analyzed (Participants) | 13 | 56 | 36
  Cough, Week 54 | 0.08 (0.89) | -0.45 (1.06) | -0.63 (1.23)
  Cough, Week 55: number analyzed (Participants) | 12 | 47 | 36
  Cough, Week 55 | 0.29 (1.05) | -0.38 (1.12) | -0.68 (1.17)
  Cough, Week 56: number analyzed (Participants) | 11 | 50 | 36
  Cough, Week 56 | 0.14 (1.05) | -0.46 (1.13) | -0.51 (1.07)
  Cough, Week 57: number analyzed (Participants) | 10 | 52 | 33
  Cough, Week 57 | 0.10 (0.81) | -0.36 (1.25) | -0.74 (1.10)
  Cough, Week 58: number analyzed (Participants) | 8 | 45 | 29
  Cough, Week 58 | 0.06 (0.94) | -0.51 (1.14) | -0.67 (1.06)
  Cough, Week 59: number analyzed (Participants) | 11 | 47 | 27
  Cough, Week 59 | 0.18 (0.81) | -0.45 (1.19) | -0.81 (1.12)
  Cough, Week 60: number analyzed (Participants) | 11 | 41 | 31
  Cough, Week 60 | 0.14 (0.71) | -0.41 (1.26) | -0.69 (1.04)
  Cough, Week 61: number analyzed (Participants) | 9 | 40 | 28
  Cough, Week 61 | 0.00 (0.97) | -0.38 (1.27) | -0.84 (1.08)
  Cough, Week 62: number analyzed (Participants) | 10 | 39 | 25
  Cough, Week 62 | -0.05 (0.86) | -0.29 (1.29) | -0.78 (1.04)
  Cough, Week 63: number analyzed (Participants) | 8 | 42 | 22
  Cough, Week 63 | 0.19 (0.70) | -0.30 (1.09) | -0.82 (0.99)
  Cough, Week 64: number analyzed (Participants) | 8 | 42 | 18
  Cough, Week 64 | 0.13 (1.16) | -0.27 (1.21) | -0.81 (0.93)
  Cough, Week 65: number analyzed (Participants) | 6 | 39 | 20
  Cough, Week 65 | 0.08 (0.97) | -0.28 (1.26) | -0.70 (1.15)
  Cough, Week 66: number analyzed (Participants) | 6 | 37 | 19
  Cough, Week 66 | 0.08 (0.86) | -0.30 (1.22) | -0.82 (1.15)
  Cough, Week 67: number analyzed (Participants) | 5 | 33 | 20
  Cough, Week 67 | -0.30 (0.67) | -0.44 (1.29) | -0.78 (1.09)
  Cough, Week 68: number analyzed (Participants) | 6 | 33 | 19
  Cough, Week 68 | 0.00 (0.95) | -0.21 (1.36) | -0.66 (1.17)
  Cough, Week 69: number analyzed (Participants) | 5 | 31 | 18
  Cough, Week 69 | 0.20 (0.91) | -0.26 (1.29) | -0.78 (1.14)
  Cough, Week 70: number analyzed (Participants) | 5 | 32 | 19
  Cough, Week 70 | 0.20 (0.91) | -0.28 (1.13) | -0.92 (1.18)
  Cough, Week 71: number analyzed (Participants) | 6 | 27 | 15
  Cough, Week 71 | -0.17 (1.21) | -0.15 (1.01) | -0.90 (1.21)
  Cough, Week 72: number analyzed (Participants) | 9 | 27 | 18
  Cough, Week 72 | 0.00 (1.38) | -0.19 (1.10) | -0.72 (1.05)
  Cough, Week 73: number analyzed (Participants) | 6 | 27 | 13
  Cough, Week 73 | 0.00 (1.38) | -0.22 (1.15) | -1.00 (1.38)
  Cough, Week 74: number analyzed (Participants) | 7 | 29 | 12
  Cough, Week 74 | 0.07 (0.89) | -0.22 (0.97) | -1.04 (1.21)
  Cough, Week 75: number analyzed (Participants) | 6 | 24 | 12
  Cough, Week 75 | 0.08 (1.24) | -0.17 (1.12) | -1.04 (1.29)
  Cough, Week 76: number analyzed (Participants) | 6 | 23 | 14
  Cough, Week 76 | 0.00 (1.38) | 0.07 (1.16) | -1.18 (1.12)
  Cough, Week 77: number analyzed (Participants) | 6 | 22 | 10
  Cough, Week 77 | 0.25 (1.29) | -0.18 (1.29) | -0.60 (1.05)
  Cough, Week 78: number analyzed (Participants) | 7 | 22 | 11
  Cough, Week 78 | 0.00 (1.26) | -0.30 (1.08) | -0.86 (1.12)
  Cough, Week 79: number analyzed (Participants) | 6 | 24 | 9
  Cough, Week 79 | 0.00 (1.38) | -0.04 (1.04) | -0.61 (1.41)
  Cough, Week 80: number analyzed (Participants) | 7 | 20 | 11
  Cough, Week 80 | 0.21 (1.07) | -0.45 (1.17) | -0.95 (1.13)
  Cough, Week 81: number analyzed (Participants) | 6 | 18 | 9
  Cough, Week 81 | 0.08 (1.02) | -0.31 (1.14) | -0.72 (1.25)
  Cough, Week 82: number analyzed (Participants) | 7 | 21 | 9
  Cough, Week 82 | 0.43 (1.17) | -0.33 (1.06) | -0.44 (1.13)
  Cough, Week 83: number analyzed (Participants) | 5 | 19 | 10
  Cough, Week 83 | 0.30 (1.44) | -0.39 (1.06) | -1.00 (1.20)
  Cough, Week 84: number analyzed (Participants) | 5 | 15 | 10
  Cough, Week 84 | 0.20 (1.30) | -0.10 (1.28) | -0.90 (1.26)
  Cough, Week 85: number analyzed (Participants) | 4 | 17 | 10
  Cough, Week 85 | 1.00 (0.58) | -0.24 (1.13) | -0.60 (1.60)
  Cough, Week 86: number analyzed (Participants) | 3 | 15 | 6
  Cough, Week 86 | 1.17 (0.58) | -0.27 (1.28) | -0.42 (1.32)
  Cough, Week 87: number analyzed (Participants) | 3 | 12 | 8
  Cough, Week 87 | 0.83 (0.58) | 0.00 (1.30) | -0.94 (1.35)
  Cough, Week 88: number analyzed (Participants) | 3 | 15 | 7
  Cough, Week 88 | 0.67 (0.76) | -0.37 (1.19) | -1.29 (1.41)
  Cough, Week 89: number analyzed (Participants) | 3 | 14 | 7
  Cough, Week 89 | 0.83 (0.58) | -0.29 (1.17) | -1.14 (1.31)
  Cough, Week 90: number analyzed (Participants) | 3 | 13 | 7
  Cough, Week 90 | 1.00 (0.50) | -0.35 (1.14) | -0.79 (1.29)
  Cough, Week 91: number analyzed (Participants) | 3 | 13 | 7
  Cough, Week 91 | 0.67 (0.76) | -0.58 (1.19) | -0.93 (1.37)
  Cough, Week 92: number analyzed (Participants) | 4 | 13 | 8
  Cough, Week 92 | 1.00 (0.58) | -0.19 (1.18) | -0.94 (1.37)
  Cough, Week 93: number analyzed (Participants) | 2 | 13 | 10
  Cough, Week 93 | 1.00 (0.71) | -0.42 (1.26) | -0.90 (1.13)
  Cough, Week 94: number analyzed (Participants) | 3 | 11 | 8
  Cough, Week 94 | 0.83 (0.58) | -0.41 (1.26) | -0.88 (1.25)
  Cough, Week 95: number analyzed (Participants) | 3 | 11 | 8
  Cough, Week 95 | 0.83 (0.58) | 0.00 (1.28) | -0.81 (1.31)
  Cough, Week 96: number analyzed (Participants) | 3 | 11 | 8
  Cough, Week 96 | 0.83 (0.58) | -0.18 (1.45) | -1.00 (1.31)
  Cough, Week 97: number analyzed (Participants) | 3 | 11 | 9
  Cough, Week 97 | 1.00 (0.50) | -0.14 (1.12) | -0.78 (1.23)
  Cough, Week 98: number analyzed (Participants) | 3 | 10 | 7
  Cough, Week 98 | 0.50 (0.50) | -0.35 (1.18) | -1.00 (1.29)
  Cough, Week 99: number analyzed (Participants) | 3 | 10 | 7
  Cough, Week 99 | 0.83 (0.58) | 0.00 (1.41) | -0.64 (1.14)
  Cough, Week 100: number analyzed (Participants) | 2 | 10 | 8
  Cough, Week 100 | 1.00 (0.71) | -0.35 (1.16) | -0.81 (1.25)
  Cough, Week 101: number analyzed (Participants) | 3 | 10 | 7
  Cough, Week 101 | 0.83 (0.58) | -0.20 (1.32) | -0.79 (1.32)
  Cough, Week 102: number analyzed (Participants) | 3 | 6 | 6
  Cough, Week 102 | 0.67 (0.76) | 0.00 (1.30) | -0.75 (1.44)
  Cough, Week 103: number analyzed (Participants) | 2 | 9 | 6
  Cough, Week 103 | 0.50 (0.00) | -0.56 (1.07) | -0.67 (1.44)
  Cough, Week 104: number analyzed (Participants) | 2 | 8 | 4
  Cough, Week 104 | 0.50 (0.00) | -0.38 (1.19) | 0.00 (1.08)
  Cough, Week 105: number analyzed (Participants) | 2 | 6 | 6
  Cough, Week 105 | 0.50 (0.00) | 0.08 (0.80) | -0.25 (1.33)
  Cough, Week 106: number analyzed (Participants) | 2 | 9 | 5
  Cough, Week 106 | 0.50 (0.00) | -0.28 (1.23) | -0.80 (1.04)
  Cough, Week 107: number analyzed (Participants) | 2 | 7 | 4
  Cough, Week 107 | 0.25 (0.35) | -0.57 (1.48) | -1.25 (1.19)
  Cough, Week 108: number analyzed (Participants) | 2 | 5 | 4
  Cough, Week 108 | 0.25 (0.35) | -0.70 (1.64) | -1.38 (1.11)
  Cough, Week 109: number analyzed (Participants) | 2 | 5 | 2
  Cough, Week 109 | 0.50 (0.00) | -0.30 (1.82) | -0.75 (1.06)
  Cough, Week 110: number analyzed (Participants) | 2 | 3 | 4
  Cough, Week 110 | 0.50 (0.00) | 0.50 (1.80) | -1.25 (1.04)
  Cough, Week 111: number analyzed (Participants) | 2 | 4 | 4
  Cough, Week 111 | 0.75 (0.35) | -0.13 (1.93) | -1.25 (1.04)
  Cough, Week 112: number analyzed (Participants) | 2 | 3 | 2
  Cough, Week 112 | 0.50 (0.00) | 0.17 (1.44) | -1.75 (0.35)
  Cough, Week 113: number analyzed (Participants) | 1 | 4 | 3
  Cough, Week 113 | 0.50 | 0.13 (1.75) | -1.17 (1.04)
  Cough, Week 114: number analyzed (Participants) | 2 | 3 | 2
  Cough, Week 114 | 0.25 (0.35) | 0.50 (1.80) | -1.50 (0.71)
  Cough, Week 115: number analyzed (Participants) | 2 | 4 | 3
  Cough, Week 115 | 0.50 (0.00) | -0.88 (1.31) | -1.00 (1.00)
  Cough, Week 116: number analyzed (Participants) | 2 | 3 | 3
  Cough, Week 116 | 0.75 (0.35) | -0.50 (1.32) | -1.33 (1.15)
  Cough, Week 117: number analyzed (Participants) | 2 | 2 | 2
  Cough, Week 117 | 0.75 (0.35) | -0.25 (1.77) | -1.50 (0.71)
  Cough, Week 118: number analyzed (Participants) | 1 | 1 | 2
  Cough, Week 118 | 0.50 | 1.00 | -1.50 (0.71)
  Cough, Week 119: number analyzed (Participants) | 0 | 1 | 2
  Cough, Week 119 |  | 1.00 | -1.00 (0.71)
  Cough, Week 120: number analyzed (Participants) | 0 | 1 | 2
  Cough, Week 120 |  | 1.00 | -1.00 (0.71)
  Cough, Week 121: number analyzed (Participants) | 0 | 1 | 2
  Cough, Week 121 |  | 1.00 | -1.00 (0.71)
  Cough, Week 122: number analyzed (Participants) | 0 | 1 | 2
  Cough, Week 122 |  | 1.00 | -1.25 (0.35)
  Cough, Week 123: number analyzed (Participants) | 0 | 1 | 1
  Cough, Week 123 |  | 1.00 | -2.00
  Cough, Week 124: number analyzed (Participants) | 0 | 1 | 1
  Cough, Week 124 |  | 2.00 | -1.00
  Cough, Week 125: number analyzed (Participants) | 0 | 0 | 1
  Cough, Week 125 |  |  | -2.00
  Cough, Week 126: number analyzed (Participants) | 0 | 0 | 1
  Cough, Week 126 |  |  | -1.00
  Cough, Week 127: number analyzed (Participants) | 0 | 0 | 1
  Cough, Week 127 |  |  | -1.00
  Cough, Time of First Pd: number analyzed (Participants) | 103 | 107 | 106
  Cough, Time of First Pd | -0.15 (1.05) | -0.16 (1.12) | -0.16 (1.05)
  Cough, Time of Last Tx Dose: number analyzed (Participants) | 161 | 172 | 151
  Cough, Time of Last Tx Dose | -0.31 (1.10) | -0.24 (1.09) | -0.21 (1.13)
  Cough, Survival Follow-Up Month 1: number analyzed (Participants) | 86 | 0 | 0
  Cough, Survival Follow-Up Month 1 | -0.03 (1.13) |  |
  Cough, Survival Follow-Up Month 2: number analyzed (Participants) | 52 | 0 | 0
  Cough, Survival Follow-Up Month 2 | 0.03 (1.04) |  |
  Cough, Survival Follow-Up Month 3: number analyzed (Participants) | 40 | 0 | 0
  Cough, Survival Follow-Up Month 3 | -0.18 (1.06) |  |
  Cough, Survival Follow-Up Month 4: number analyzed (Participants) | 32 | 0 | 0
  Cough, Survival Follow-Up Month 4 | -0.09 (1.32) |  |
  Cough, Survival Follow-Up Month 5: number analyzed (Participants) | 26 | 0 | 0
  Cough, Survival Follow-Up Month 5 | -0.04 (1.14) |  |
  Cough, Survival Follow-Up Month 6: number analyzed (Participants) | 23 | 0 | 0
  Cough, Survival Follow-Up Month 6 | -0.17 (1.17) |  |
  Cough, Survival Follow-Up Month 7: number analyzed (Participants) | 3 | 0 | 0
  Cough, Survival Follow-Up Month 7 | 1.33 (0.29) |  |
  Cough, Survival Follow-Up Month 8: number analyzed (Participants) | 2 | 0 | 0
  Cough, Survival Follow-Up Month 8 | -0.50 (2.12) |  |
  Dyspnoea, Week 1: number analyzed (Participants) | 171 | 192 | 166
  Dyspnoea, Week 1 | 0.18 (0.80) | 0.11 (0.76) | 0.17 (0.73)
  Dyspnoea, Week 2: number analyzed (Participants) | 160 | 186 | 165
  Dyspnoea, Week 2 | 0.13 (0.75) | 0.11 (0.86) | 0.27 (0.88)
  Dyspnoea, Week 3: number analyzed (Participants) | 165 | 175 | 165
  Dyspnoea, Week 3 | 0.06 (0.83) | 0.16 (0.81) | 0.30 (0.89)
  Dyspnoea, Week 4: number analyzed (Participants) | 157 | 173 | 169
  Dyspnoea, Week 4 | 0.17 (0.89) | 0.16 (0.83) | 0.26 (0.89)
  Dyspnoea, Week 5: number analyzed (Participants) | 160 | 172 | 159
  Dyspnoea, Week 5 | 0.21 (0.89) | 0.25 (0.88) | 0.31 (0.85)
  Dyspnoea, Week 6: number analyzed (Participants) | 151 | 170 | 161
  Dyspnoea, Week 6 | 0.17 (0.97) | 0.23 (0.83) | 0.29 (0.88)
  Dyspnoea, Week 7: number analyzed (Participants) | 138 | 166 | 143
  Dyspnoea, Week 7 | 0.20 (0.98) | 0.25 (0.91) | 0.27 (0.96)
  Dyspnoea, Week 8: number analyzed (Participants) | 140 | 162 | 152
  Dyspnoea, Week 8 | 0.26 (0.95) | 0.29 (0.91) | 0.31 (0.97)
  Dyspnoea, Week 9: number analyzed (Participants) | 135 | 162 | 143
  Dyspnoea, Week 9 | 0.23 (0.97) | 0.26 (0.85) | 0.33 (0.98)
  Dyspnoea, Week 10: number analyzed (Participants) | 133 | 158 | 146
  Dyspnoea, Week 10 | 0.37 (0.99) | 0.34 (0.94) | 0.34 (0.95)
  Dyspnoea, Week 11: number analyzed (Participants) | 132 | 157 | 137
  Dyspnoea, Week 11 | 0.40 (0.95) | 0.31 (0.91) | 0.35 (0.97)
  Dyspnoea, Week 12: number analyzed (Participants) | 128 | 151 | 136
  Dyspnoea, Week 12 | 0.44 (0.98) | 0.41 (1.01) | 0.29 (0.90)
  Dyspnoea, Week 13: number analyzed (Participants) | 117 | 144 | 130
  Dyspnoea, Week 13 | 0.40 (1.03) | 0.32 (0.92) | 0.34 (0.94)
  Dyspnoea, Week 14: number analyzed (Participants) | 105 | 139 | 138
  Dyspnoea, Week 14 | 0.42 (0.95) | 0.29 (0.92) | 0.34 (0.91)
  Dyspnoea, Week 15: number analyzed (Participants) | 97 | 143 | 132
  Dyspnoea, Week 15 | 0.36 (0.98) | 0.32 (0.92) | 0.30 (0.91)
  Dyspnoea, Week 16: number analyzed (Participants) | 102 | 138 | 121
  Dyspnoea, Week 16 | 0.45 (0.95) | 0.32 (0.93) | 0.36 (0.92)
  Dyspnoea, Week 17: number analyzed (Participants) | 101 | 135 | 129
  Dyspnoea, Week 17 | 0.55 (0.99) | 0.25 (0.90) | 0.29 (0.91)
  Dyspnoea, Week 18: number analyzed (Participants) | 93 | 141 | 129
  Dyspnoea, Week 18 | 0.46 (0.93) | 0.28 (0.93) | 0.34 (0.97)
  Dyspnoea, Week 19: number analyzed (Participants) | 85 | 129 | 118
  Dyspnoea, Week 19 | 0.48 (0.97) | 0.28 (0.98) | 0.44 (0.96)
  Dyspnoea, Week 20: number analyzed (Participants) | 75 | 130 | 114
  Dyspnoea, Week 20 | 0.37 (0.97) | 0.28 (0.93) | 0.24 (0.99)
  Dyspnoea, Week 21: number analyzed (Participants) | 69 | 129 | 113
  Dyspnoea, Week 21 | 0.51 (0.94) | 0.23 (0.98) | 0.19 (1.00)
  Dyspnoea, Week 22: number analyzed (Participants) | 79 | 125 | 109
  Dyspnoea, Week 22 | 0.50 (0.95) | 0.25 (0.96) | 0.24 (1.07)
  Dyspnoea, Week 23: number analyzed (Participants) | 70 | 128 | 106
  Dyspnoea, Week 23 | 0.44 (0.94) | 0.30 (0.99) | 0.20 (0.98)
  Dyspnoea, Week 24: number analyzed (Participants) | 67 | 121 | 105
  Dyspnoea, Week 24 | 0.25 (1.01) | 0.20 (0.91) | 0.29 (1.02)
  Dyspnoea, Week 25: number analyzed (Participants) | 48 | 118 | 104
  Dyspnoea, Week 25 | 0.27 (0.94) | 0.18 (0.95) | 0.25 (1.00)
  Dyspnoea, Week 26: number analyzed (Participants) | 48 | 111 | 99
  Dyspnoea, Week 26 | 0.20 (0.84) | 0.31 (0.96) | 0.39 (1.02)
  Dyspnoea, Week 27: number analyzed (Participants) | 42 | 110 | 95
  Dyspnoea, Week 27 | 0.31 (0.80) | 0.21 (0.95) | 0.36 (1.14)
  Dyspnoea, Week 28: number analyzed (Participants) | 41 | 103 | 88
  Dyspnoea, Week 28 | 0.24 (0.83) | 0.17 (0.86) | 0.30 (1.07)
  Dyspnoea, Week 29: number analyzed (Participants) | 38 | 100 | 89
  Dyspnoea, Week 29 | 0.30 (0.82) | 0.19 (0.96) | 0.31 (1.07)
  Dyspnoea, Week 30: number analyzed (Participants) | 46 | 104 | 86
  Dyspnoea, Week 30 | 0.30 (0.82) | 0.12 (0.94) | 0.39 (1.08)
  Dyspnoea, Week 31: number analyzed (Participants) | 35 | 97 | 77
  Dyspnoea, Week 31 | 0.34 (0.76) | 0.18 (0.96) | 0.36 (1.12)
  Dyspnoea, Week 32: number analyzed (Participants) | 29 | 91 | 70
  Dyspnoea, Week 32 | 0.28 (0.79) | 0.09 (0.84) | 0.26 (1.05)
  Dyspnoea, Week 33: number analyzed (Participants) | 29 | 93 | 68
  Dyspnoea, Week 33 | 0.39 (0.74) | 0.02 (0.85) | 0.31 (1.05)
  Dyspnoea, Week 34: number analyzed (Participants) | 33 | 92 | 73
  Dyspnoea, Week 34 | 0.32 (0.69) | 0.05 (0.76) | 0.30 (1.05)
  Dyspnoea, Week 35: number analyzed (Participants) | 33 | 90 | 72
  Dyspnoea, Week 35 | 0.35 (0.88) | 0.04 (0.82) | 0.38 (1.05)
  Dyspnoea, Week 36: number analyzed (Participants) | 31 | 83 | 64
  Dyspnoea, Week 36 | 0.32 (0.68) | 0.11 (0.82) | 0.37 (0.98)
  Dyspnoea, Week 37: number analyzed (Participants) | 24 | 84 | 65
  Dyspnoea, Week 37 | 0.24 (0.76) | 0.16 (0.92) | 0.32 (0.92)
  Dyspnoea, Week 38: number analyzed (Participants) | 24 | 86 | 65
  Dyspnoea, Week 38 | 0.31 (0.75) | 0.10 (0.78) | 0.40 (1.01)
  Dyspnoea, Week 39: number analyzed (Participants) | 25 | 75 | 68
  Dyspnoea, Week 39 | 0.39 (0.76) | 0.04 (0.87) | 0.36 (1.01)
  Dyspnoea, Week 40: number analyzed (Participants) | 24 | 74 | 62
  Dyspnoea, Week 40 | 0.38 (0.74) | 0.24 (0.92) | 0.37 (0.91)
  Dyspnoea, Week 41: number analyzed (Participants) | 22 | 69 | 60
  Dyspnoea, Week 41 | 0.45 (0.92) | 0.13 (0.84) | 0.33 (0.89)
  Dyspnoea, Week 42: number analyzed (Participants) | 24 | 77 | 60
  Dyspnoea, Week 42 | 0.37 (0.82) | 0.05 (0.81) | 0.29 (1.02)
  Dyspnoea, Week 43: number analyzed (Participants) | 23 | 72 | 58
  Dyspnoea, Week 43 | 0.48 (0.94) | 0.16 (0.76) | 0.41 (1.05)
  Dyspnoea, Week 44: number analyzed (Participants) | 20 | 63 | 60
  Dyspnoea, Week 44 | 0.22 (0.95) | 0.11 (0.88) | 0.33 (1.08)
  Dyspnoea, Week 45: number analyzed (Participants) | 20 | 64 | 51
  Dyspnoea, Week 45 | 0.32 (1.04) | 0.20 (0.84) | 0.27 (1.07)
  Dyspnoea, Week 46: number analyzed (Participants) | 20 | 61 | 53
  Dyspnoea, Week 46 | 0.36 (0.98) | 0.08 (0.78) | 0.26 (0.99)
  Dyspnoea, Week 47: number analyzed (Participants) | 20 | 64 | 48
  Dyspnoea, Week 47 | 0.32 (0.85) | 0.06 (0.80) | 0.31 (1.01)
  Dyspnoea, Week 48: number analyzed (Participants) | 19 | 62 | 52
  Dyspnoea, Week 48 | 0.32 (0.88) | 0.14 (0.85) | 0.22 (0.93)
  Dyspnoea, Week 49: number analyzed (Participants) | 13 | 57 | 45
  Dyspnoea, Week 49 | 0.46 (0.99) | 0.06 (0.78) | 0.14 (0.93)
  Dyspnoea, Week 50: number analyzed (Participants) | 15 | 60 | 45
  Dyspnoea, Week 50 | 0.41 (0.84) | 0.10 (0.85) | 0.06 (0.86)
  Dyspnoea, Week 51: number analyzed (Participants) | 11 | 58 | 37
  Dyspnoea, Week 51 | 0.71 (0.92) | 0.08 (0.78) | 0.15 (1.06)
  Dyspnoea, Week 52: number analyzed (Participants) | 13 | 58 | 43
  Dyspnoea, Week 52 | 0.60 (0.81) | 0.11 (0.86) | 0.34 (0.97)
  Dyspnoea, Week 53: number analyzed (Participants) | 14 | 53 | 35
  Dyspnoea, Week 53 | 0.70 (0.85) | 0.11 (0.89) | 0.11 (1.11)
  Dyspnoea, Week 54: number analyzed (Participants) | 13 | 56 | 36
  Dyspnoea, Week 54 | 0.71 (0.94) | 0.11 (0.80) | 0.10 (1.02)
  Dyspnoea, Week 55: number analyzed (Participants) | 12 | 47 | 36
  Dyspnoea, Week 55 | 0.82 (0.93) | 0.15 (0.85) | 0.16 (1.08)
  Dyspnoea, Week 56: number analyzed (Participants) | 11 | 50 | 36
  Dyspnoea, Week 56 | 0.69 (0.94) | 0.14 (0.95) | 0.12 (1.02)
  Dyspnoea, Week 57: number analyzed (Participants) | 10 | 52 | 33
  Dyspnoea, Week 57 | 0.74 (0.80) | 0.12 (0.90) | 0.13 (1.03)
  Dyspnoea, Week 58: number analyzed (Participants) | 8 | 45 | 29
  Dyspnoea, Week 58 | 0.80 (0.93) | 0.02 (0.98) | 0.12 (1.06)
  Dyspnoea, Week 59: number analyzed (Participants) | 11 | 47 | 27
  Dyspnoea, Week 59 | 0.78 (1.09) | 0.11 (1.00) | -0.03 (1.04)
  Dyspnoea, Week 60: number analyzed (Participants) | 11 | 41 | 31
  Dyspnoea, Week 60 | 0.67 (0.86) | 0.06 (0.93) | 0.02 (1.02)
  Dyspnoea, Week 61: number analyzed (Participants) | 9 | 40 | 28
  Dyspnoea, Week 61 | 0.91 (0.91) | 0.05 (0.92) | -0.18 (0.93)
  Dyspnoea, Week 62: number analyzed (Participants) | 10 | 39 | 25
  Dyspnoea, Week 62 | 0.58 (0.94) | 0.01 (0.96) | -0.04 (1.01)
  Dyspnoea, Week 63: number analyzed (Participants) | 8 | 42 | 22
  Dyspnoea, Week 63 | 0.58 (1.14) | 0.10 (0.95) | -0.06 (0.72)
  Dyspnoea, Week 64: number analyzed (Participants) | 8 | 42 | 18
  Dyspnoea, Week 64 | 0.63 (0.98) | 0.07 (1.08) | -0.22 (0.74)
  Dyspnoea, Week 65: number analyzed (Participants) | 6 | 39 | 20
  Dyspnoea, Week 65 | 0.80 (1.06) | 0.05 (1.05) | -0.18 (0.87)
  Dyspnoea, Week 66: number analyzed (Participants) | 6 | 37 | 19
  Dyspnoea, Week 66 | 0.70 (1.02) | 0.04 (1.07) | -0.18 (0.85)
  Dyspnoea, Week 67: number analyzed (Participants) | 5 | 33 | 20
  Dyspnoea, Week 67 | 0.52 (0.95) | 0.04 (1.15) | -0.24 (0.97)
  Dyspnoea, Week 68: number analyzed (Participants) | 6 | 33 | 19
  Dyspnoea, Week 68 | 0.63 (0.98) | 0.01 (1.07) | -0.11 (0.86)
  Dyspnoea, Week 69: number analyzed (Participants) | 5 | 31 | 18
  Dyspnoea, Week 69 | 0.96 (0.59) | 0.06 (1.19) | -0.20 (0.87)
  Dyspnoea, Week 70: number analyzed (Participants) | 5 | 32 | 19
  Dyspnoea, Week 70 | 1.00 (0.60) | 0.16 (1.08) | -0.18 (0.94)
  Dyspnoea, Week 71: number analyzed (Participants) | 6 | 27 | 15
  Dyspnoea, Week 71 | 0.70 (0.91) | 0.22 (1.08) | -0.01 (0.82)
  Dyspnoea, Week 72: number analyzed (Participants) | 6 | 27 | 18
  Dyspnoea, Week 72 | 0.57 (0.98) | 0.25 (1.16) | -0.06 (0.79)
  Dyspnoea, Week 73: number analyzed (Participants) | 6 | 27 | 13
  Dyspnoea, Week 73 | 0.67 (1.07) | 0.10 (1.18) | -0.11 (0.79)
  Dyspnoea, Week 74: number analyzed (Participants) | 7 | 29 | 12
  Dyspnoea, Week 74 | 0.74 (0.96) | 0.10 (1.15) | -0.17 (0.86)
  Dyspnoea, Week 75: number analyzed (Participants) | 6 | 24 | 12
  Dyspnoea, Week 75 | 0.70 (0.99) | 0.05 (1.13) | -0.22 (0.81)
  Dyspnoea, Week 76: number analyzed (Participants) | 6 | 23 | 14
  Dyspnoea, Week 76 | 0.67 (0.90) | 0.25 (1.33) | -0.13 (0.90)
  Dyspnoea, Week 77: number analyzed (Participants) | 6 | 22 | 10
  Dyspnoea, Week 77 | 0.73 (0.95) | 0.04 (1.36) | 0.12 (0.76)
  Dyspnoea, Week 78: number analyzed (Participants) | 7 | 22 | 11
  Dyspnoea, Week 78 | 0.57 (0.94) | 0.09 (1.24) | -0.20 (0.95)
  Dyspnoea, Week 79: number analyzed (Participants) | 6 | 24 | 9
  Dyspnoea, Week 79 | 0.57 (0.77) | 0.16 (1.29) | -0.13 (0.93)
  Dyspnoea, Week 80: number analyzed (Participants) | 7 | 20 | 11
  Dyspnoea, Week 80 | 0.60 (0.78) | -0.13 (1.17) | 0.00 (0.81)
  Dyspnoea, Week 81: number analyzed (Participants) | 6 | 18 | 9
  Dyspnoea, Week 81 | 0.50 (0.92) | -0.02 (1.17) | -0.04 (0.86)
  Dyspnoea, Week 82: number analyzed (Participants) | 7 | 21 | 9
  Dyspnoea, Week 82 | 0.57 (0.91) | -0.05 (1.16) | 0.00 (0.90)
  Dyspnoea, Week 83: number analyzed (Participants) | 5 | 19 | 10
  Dyspnoea, Week 83 | 0.28 (0.69) | -0.08 (1.26) | -0.40 (0.98)
  Dyspnoea, Week 84: number analyzed (Participants) | 5 | 15 | 10
  Dyspnoea, Week 84 | 0.16 (0.59) | -0.17 (1.23) | -0.22 (0.99)
  Dyspnoea, Week 85: number analyzed (Participants) | 4 | 17 | 10
  Dyspnoea, Week 85 | 0.70 (0.50) | -0.16 (1.11) | -0.16 (1.03)
  Dyspnoea, Week 86: number analyzed (Participants) | 3 | 15 | 6
  Dyspnoea, Week 86 | 1.33 (1.45) | -0.23 (1.12) | -0.17 (1.26)
  Dyspnoea, Week 87: number analyzed (Participants) | 3 | 12 | 8
  Dyspnoea, Week 87 | 0.40 (0.40) | 0.08 (1.45) | -0.25 (1.06)
  Dyspnoea, Week 88: number analyzed (Participants) | 3 | 15 | 7
  Dyspnoea, Week 88 | 0.40 (0.69) | -0.21 (1.06) | -0.51 (1.06)
  Dyspnoea, Week 89: number analyzed (Participants) | 3 | 14 | 7
  Dyspnoea, Week 89 | 0.53 (0.42) | -0.13 (1.02) | -0.06 (1.12)
  Dyspnoea, Week 90: number analyzed (Participants) | 3 | 13 | 7
  Dyspnoea, Week 90 | 0.27 (0.31) | -0.32 (0.99) | -0.17 (1.07)
  Dyspnoea, Week 91: number analyzed (Participants) | 3 | 13 | 7
  Dyspnoea, Week 91 | 0.33 (0.31) | -0.52 (0.81) | -0.17 (1.13)
  Dyspnoea, Week 92: number analyzed (Participants) | 4 | 13 | 8
  Dyspnoea, Week 92 | 0.75 (0.66) | -0.28 (1.02) | -0.10 (1.06)
  Dyspnoea, Week 93: number analyzed (Participants) | 2 | 13 | 10
  Dyspnoea, Week 93 | 0.40 (0.28) | -0.23 (0.93) | -0.14 (0.90)
  Dyspnoea, Week 94: number analyzed (Participants) | 3 | 11 | 8
  Dyspnoea, Week 94 | 0.67 (0.70) | -0.38 (0.85) | -0.25 (0.98)
  Dyspnoea, Week 95: number analyzed (Participants) | 3 | 11 | 8
  Dyspnoea, Week 95 | 0.53 (0.23) | -0.07 (1.21) | -0.20 (1.04)
  Dyspnoea, Week 96: number analyzed (Participants) | 3 | 11 | 8
  Dyspnoea, Week 96 | 0.33 (0.42) | -0.02 (1.21) | -0.18 (1.09)
  Dyspnoea, Week 97: number analyzed (Participants) | 3 | 11 | 9
  Dyspnoea, Week 97 | 0.67 (0.42) | -0.22 (1.18) | 0.04 (1.13)
  Dyspnoea, Week 98: number analyzed (Participants) | 3 | 10 | 7
  Dyspnoea, Week 98 | 0.73 (0.50) | -0.18 (1.19) | -0.29 (1.08)
  Dyspnoea, Week 99: number analyzed (Participants) | 3 | 10 | 7
  Dyspnoea, Week 99 | 0.47 (0.46) | -0.26 (1.25) | -0.29 (1.09)
  Dyspnoea, Week 100: number analyzed (Participants) | 2 | 10 | 8
  Dyspnoea, Week 100 | 0.50 (0.42) | -0.24 (1.24) | -0.20 (1.08)
  Dyspnoea, Week 101: number analyzed (Participants) | 3 | 10 | 7
  Dyspnoea, Week 101 | 0.40 (0.35) | -0.26 (1.23) | -0.03 (1.09)
  Dyspnoea, Week 102: number analyzed (Participants) | 3 | 6 | 6
  Dyspnoea, Week 102 | 0.40 (0.35) | -0.67 (0.89) | 0.00 (1.08)
  Dyspnoea, Week 103: number analyzed (Participants) | 2 | 9 | 6
  Dyspnoea, Week 103 | 0.70 (0.42) | -0.60 (0.73) | -0.03 (1.24)
  Dyspnoea, Week 104: number analyzed (Participants) | 2 | 8 | 4
  Dyspnoea, Week 104 | 0.50 (0.71) | -0.63 (0.82) | -0.35 (1.42)
  Dyspnoea, Week 105: number analyzed (Participants) | 2 | 6 | 6
  Dyspnoea, Week 105 | 0.40 (0.57) | -0.20 (0.33) | 0.23 (0.92)
  Dyspnoea, Week 106: number analyzed (Participants) | 2 | 9 | 5
  Dyspnoea, Week 106 | 0.30 (0.42) | -0.24 (0.31) | -0.04 (0.57)
  Dyspnoea, Week 107: number analyzed (Participants) | 2 | 7 | 4
  Dyspnoea, Week 107 | 0.60 (0.28) | -0.17 (0.35) | -0.30 (0.74)
  Dyspnoea, Week 108: number analyzed (Participants) | 2 | 5 | 4
  Dyspnoea, Week 108 | 0.60 (0.28) | -0.36 (0.43) | -0.40 (0.88)
  Dyspnoea, Week 109: number analyzed (Participants) | 2 | 5 | 2
  Dyspnoea, Week 109 | 0.80 (0.00) | -0.40 (0.47) | 0.10 (0.99)
  Dyspnoea, Week 110: number analyzed (Participants) | 2 | 3 | 4
  Dyspnoea, Week 110 | 0.60 (0.28) | -0.27 (0.50) | -0.40 (0.94)
  Dyspnoea, Week 111: number analyzed (Participants) | 2 | 4 | 4
  Dyspnoea, Week 111 | 0.30 (0.42) | -0.15 (0.34) | -0.45 (0.91)
  Dyspnoea, Week 112: number analyzed (Participants) | 2 | 3 | 2
  Dyspnoea, Week 112 | 0.50 (0.42) | -0.20 (0.40) | -1.30 (0.14)
  Dyspnoea, Week 113: number analyzed (Participants) | 1 | 4 | 3
  Dyspnoea, Week 113 | 1.00 | -0.35 (0.44) | -0.47 (1.14)
  Dyspnoea, Week 114: number analyzed (Participants) | 2 | 3 | 2
  Dyspnoea, Week 114 | 0.50 (0.71) | -0.27 (0.50) | -1.30 (0.14)
  Dyspnoea, Week 115: number analyzed (Participants) | 2 | 4 | 3
  Dyspnoea, Week 115 | 0.50 (0.71) | -0.40 (0.28) | -0.67 (1.10)
  Dyspnoea, Week 116: number analyzed (Participants) | 2 | 3 | 3
  Dyspnoea, Week 116 | 0.40 (0.57) | -0.20 (0.53) | -0.73 (1.17)
  Dyspnoea, Week 117: number analyzed (Participants) | 2 | 2 | 2
  Dyspnoea, Week 117 | 0.40 (0.28) | -0.60 (0.28) | -1.20 (0.28)
  Dyspnoea, Week 118: number analyzed (Participants) | 1 | 1 | 2
  Dyspnoea, Week 118 | 1.00 | -0.80 | -1.20 (0.57)
  Dyspnoea, Week 119: number analyzed (Participants) | 0 | 1 | 2
  Dyspnoea, Week 119 |  | -0.80 | -1.40 (0.28)
  Dyspnoea, Week 120: number analyzed (Participants) | 0 | 1 | 2
  Dyspnoea, Week 120 |  | -0.80 | -1.10 (0.42)
  Dyspnoea, Week 121: number analyzed (Participants) | 0 | 1 | 2
  Dyspnoea, Week 121 |  | -0.80 | -1.30 (0.14)
  Dyspnoea, Week 122: number analyzed (Participants) | 0 | 1 | 2
  Dyspnoea, Week 122 |  | -0.80 | -1.30 (0.14)
  Dyspnoea, Week 123: number analyzed (Participants) | 0 | 1 | 1
  Dyspnoea, Week 123 |  | -0.80 | -1.00
  Dyspnoea, Week 124: number analyzed (Participants) | 0 | 1 | 1
  Dyspnoea, Week 124 |  | -0.80 | -1.20
  Dyspnoea, Week 125: number analyzed (Participants) | 0 | 0 | 1
  Dyspnoea, Week 125 |  |  | -1.00
  Dyspnoea, Week 126: number analyzed (Participants) | 0 | 0 | 1
  Dyspnoea, Week 126 |  |  | -1.20
  Dyspnoea, Week 127: number analyzed (Participants) | 0 | 0 | 1
  Dyspnoea, Week 127 |  |  | -1.20
  Dyspnoea, Time of First Pd: number analyzed (Participants) | 103 | 107 | 106
  Dyspnoea, Time of First Pd | 0.38 (1.06) | 0.42 (0.95) | 0.27 (1.13)
  Dyspnoea, Time of Last Tx Dose: number analyzed (Participants) | 161 | 172 | 151
  Dyspnoea, Time of Last Tx Dose | 0.43 (0.91) | 0.28 (1.01) | 0.28 (1.00)
  Dyspnoea, Survival Follow-Up Month 1: number analyzed (Participants) | 86 | 0 | 0
  Dyspnoea, Survival Follow-Up Month 1 | 0.56 (1.09) |  |
  Dyspnoea, Survival Follow-Up Month 2: number analyzed (Participants) | 52 | 0 | 0
  Dyspnoea, Survival Follow-Up Month 2 | 0.71 (0.89) |  |
  Dyspnoea, Survival Follow-Up Month 3: number analyzed (Participants) | 40 | 0 | 0
  Dyspnoea, Survival Follow-Up Month 3 | 0.67 (1.06) |  |
  Dyspnoea, Survival Follow-Up Month 4: number analyzed (Participants) | 32 | 0 | 0
  Dyspnoea, Survival Follow-Up Month 4 | 0.57 (0.91) |  |
  Dyspnoea, Survival Follow-Up Month 5: number analyzed (Participants) | 26 | 0 | 0
  Dyspnoea, Survival Follow-Up Month 5 | 0.66 (1.02) |  |
  Dyspnoea, Survival Follow-Up Month 6: number analyzed (Participants) | 23 | 0 | 0
  Dyspnoea, Survival Follow-Up Month 6 | 0.63 (1.09) |  |
  Dyspnoea, Survival Follow-Up Month 7: number analyzed (Participants) | 3 | 0 | 0
  Dyspnoea, Survival Follow-Up Month 7 | 1.07 (1.36) |  |
  Dyspnoea, Survival Follow-Up Month 8: number analyzed (Participants) | 2 | 0 | 0
  Dyspnoea, Survival Follow-Up Month 8 | 0.10 (0.14) |  |

15. Secondary Outcome: PFS as Determined by the Investigator Using RECIST v1.1 in the ITT Population (Arm A and Arm B)
Description: PFS is defined as the time between the date of randomization and the date of first documented disease progression or death, whichever occurs first, in the ITT Population Arm A and Arm B.
Time Frame: Up to approximately 30 months after first participant enrolled
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 343 | 338
Months | 6.5 [5.7 to 7.1] | 5.6 [5.5 to 6.9]
Statistical Analysis 1: Comparison: Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin vs Arm A: Atezolizumab + Paclitaxel + Carboplatin; Test type: Superiority — Stratified Analysis; p = 0.4007, Log Rank; Hazard Ratio (HR) = 0.930, 95% CI 2-sided [0.784 to 1.102]

16. Secondary Outcome: OS in the ITT Population (Arm A and Arm B)
Description: OS is defined as the time between the date of randomization and date of death from any cause in the ITT Population, Arm A and Arm B.
Time Frame: Up to approximately 39 months after first participant enrolled
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 343 | 338
Months | 14.2 [12.3 to 16.8] | 12.6 [11.6 to 14.7]

17. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Percentage of participants with at least one adverse event.
Time Frame: Up to approximately 68 months after first participant enrolled
Population: The safety population included all treated patients, defined as randomized patients who received any protocol treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm C: Nab-Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 334 | 334 | 332
Percentage of participants | 97.0 | 99.4 | 97.9

18. Secondary Outcome: Percentage of Participants With Anti-therapeutic Antibody (ATA) Response to Atezolizumab
Description: Percentage of participants with Anti-therapeutic Antibody (ATA) response to atezolizumab.
Time Frame: Up to approximately 30 months after first participant enrolled
Population: The baseline ADA evaluable population for each study treatment included participants who had a baseline ADA result. The post-baseline ADA evaluable population for each study treatment included participants who had at least one post baseline ADA result and who had received at least one dose of that study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Atezolizumab + Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin
Number analyzed (Participants) | 338 | 343
Percentage of participants
  Baseline evaluable participants: number analyzed (Participants) | 321 | 320
  Baseline evaluable participants | 3.1 | 1.9
  Post-baseline evaluable participants: number analyzed (Participants) | 308 | 313
  Post-baseline evaluable participants | 48.1 | 21.4

19. Secondary Outcome: Maximum Observed Serum Atezolizumab Concentration (Cmax)
Description: Maximum observed serum atezolizumab concentration (Cmax). The predose samples will be collected on the same day of treatment administration. The infusion duration of atezolizumab will be of 30-60 minutes.
Time Frame: Cycle 1 Day 1 and Cycle 3 Day 1 (Cycle length = 21 days)
Population: The pharmacokinetic evaluable population is defined as all participants who received any dose of atezolizumab, carboplatin, paclitaxel, or nab paclitaxel and who had evaluable PK samples post-dose.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Arm A: Atezolizumab + Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin
Number analyzed (Participants) | 327 | 328
µg/mL
  Cycle 1 Day 1 Post dose: number analyzed (Participants) | 309 | 302
  Cycle 1 Day 1 Post dose | 372 (116) | 378 (124)
  Cycle 3 Day 1 Post dose: number analyzed (Participants) | 251 | 263
  Cycle 3 Day 1 Post dose | 470 (147) | 444 (119)

20. Secondary Outcome: Minimum Observed Serum Atezolizumab Concentration (Cmin)
Description: Minimum observed serum atezolizumab concentration (Cmin). The predose samples will be collected on the same day of treatment administration.
Time Frame: Predose on Day 1 of Cycles 1-4, 8, 16, every 8 cycle thereafter (up to 30 months), at treatment discontinuation (up to 30 months), and at 120 days after the last dose of atezolizumab (up to approximately 30 months, each cycle is 21 days)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Arm A: Atezolizumab + Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin
Number analyzed (Participants) | 327 | 328
µg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 311 | 308
  Cycle 1 Day 1 | NA (NA) — Below the level of detection. | NA (NA) — Below the level of detection.
  Cycle 2 Day 1: number analyzed (Participants) | 285 | 289
  Cycle 2 Day 1 | 63.9 (29.9) | 69.5 (34.7)
  Cycle 3 Day 1: number analyzed (Participants) | 267 | 281
  Cycle 3 Day 1 | 103 (40.1) | 107 (52.0)
  Cycle 4 Day 1: number analyzed (Participants) | 256 | 252
  Cycle 4 Day 1 | 128 (62.3) | 126 (68.4)
  Cycle 8 Day 1: number analyzed (Participants) | 172 | 180
  Cycle 8 Day 1 | 188 (80.4) | 190 (84.6)
  Cycle 16 Day 1: number analyzed (Participants) | 66 | 78
  Cycle 16 Day 1 | 201 (79.2) | 212 (78.1)
  Cycle 24 Day 1: number analyzed (Participants) | 27 | 30
  Cycle 24 Day 1 | 187 (90.4) | 224 (134)
  Cycle 32 Day 1: number analyzed (Participants) | 13 | 9
  Cycle 32 Day 1 | 242 (88.4) | 210 (102)
  Cycle 40 Day 1: number analyzed (Participants) | 3 | 1
  Cycle 40 Day 1 | 308 (141) | 174 (NA) — Not evaluable; only 1 participant.
  Treatment Discontinuation Visit: number analyzed (Participants) | 133 | 140
  Treatment Discontinuation Visit | 126 (93.7) | 137 (103)
  Day 120 Post Last Dose: number analyzed (Participants) | 49 | 62
  Day 120 Post Last Dose | 7.81 (9.76) | 9.47 (13.1)

21. Secondary Outcome: Plasma Concentrations for Paclitaxel
Description: Plasma concentrations for paclitaxel.
Time Frame: Prior to infusion (within same day of treatment administration), 5-10 minutes before the end of infusion, and 1 hour after the end of infusion (infusion duration 180 minutes) on Day 1 of Cycles 1 and 3 (each cycle is 21 days)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A: Atezolizumab + Paclitaxel + Carboplatin
Number analyzed (Participants) | 35
ng/mL
  Cycle 1 Day 1 Prior to Infusion: number analyzed (Participants) | 32
  Cycle 1 Day 1 Prior to Infusion | NA (NA) — Below the level of detection.
  Cycle 1 Day 1 Before end of Infusion: number analyzed (Participants) | 30
  Cycle 1 Day 1 Before end of Infusion | 5860 (2410)
  Cycle 1 Day 1 After Infusion: number analyzed (Participants) | 33
  Cycle 1 Day 1 After Infusion | 2960 (2770)
  Cycle 3 Day 1 Prior to Infusion: number analyzed (Participants) | 24
  Cycle 3 Day 1 Prior to Infusion | NA (NA) — Below the threshold of the assay.
  Cycle 3 Day 1 Before end of Infusion: number analyzed (Participants) | 23
  Cycle 3 Day 1 Before end of Infusion | 21900 (42600)
  Cycle 3 Day 1 After Infusion: number analyzed (Participants) | 24
  Cycle 3 Day 1 After Infusion | 11000 (30700)

22. Secondary Outcome: Plasma Concentrations for Nab-Paclitaxel
Description: Plasma concentrations for nab-paclitaxel.
Time Frame: Prior to infusion (within same day of treatment administration), 5-10 minutes before the end of infusion, and 1 hour after the end of infusion (infusion duration 30 minutes) on Day 1 of Cycles 1 and 3 (each cycle is 21 days)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm C: Nab-Paclitaxel + Carboplatin
Number analyzed (Participants) | 32 | 38
ng/mL
  Cycle 1 Day 1 Prior to Infusion: number analyzed (Participants) | 26 | 37
  Cycle 1 Day 1 Prior to Infusion | NA (NA) — Below the level of detection. | NA (NA) — Below the level of detection.
  Cycle 1 Day 1 Before End of Infusion: number analyzed (Participants) | 25 | 33
  Cycle 1 Day 1 Before End of Infusion | 3330 (3680) | 8160 (20900)
  Cycle 1 Day 1 After Infusion: number analyzed (Participants) | 28 | 36
  Cycle 1 Day 1 After Infusion | 735 (1300) | 921 (2080)
  Cycle 3 Day 1 Prior to Infusion: number analyzed (Participants) | 24 | 28
  Cycle 3 Day 1 Prior to Infusion | NA (NA) — Below the threshold of the assay. | NA (NA) — Below the threshold of the assay.
  Cycle 3 Day 1 Before End of Infusion: number analyzed (Participants) | 23 | 27
  Cycle 3 Day 1 Before End of Infusion | 7160 (12300) | 7180 (14400)
  Cycle 3 Day 1 After Infusion: number analyzed (Participants) | 25 | 28
  Cycle 3 Day 1 After Infusion | 296 (274) | 1140 (2070)

23. Secondary Outcome: Plasma Concentrations for Carboplatin
Description: Plasma concentrations for carboplatin.
Time Frame: Prior to infusion (within same day of treatment administration), 5-10 minutes before the end of infusion, and 1 hour after the end of infusion (infusion duration 15 to 30 minutes) on Day 1 of Cycles 1 and 3 (each cycle is 21 days)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A: Atezolizumab + Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm C: Nab-Paclitaxel + Carboplatin
Number analyzed (Participants) | 34 | 33 | 39
ng/mL
  Cycle 1 Day 1 Prior to Infusion: number analyzed (Participants) | 31 | 29 | 34
  Cycle 1 Day 1 Prior to Infusion | NA (NA) — Below the level of detection. | NA (NA) — Below the level of detection. | NA (NA) — Below the level of detection.
  Cycle 1 Day 1 Before End of Infusion: number analyzed (Participants) | 31 | 27 | 36
  Cycle 1 Day 1 Before End of Infusion | 21100 (12400) | 15900 (9270) | 24900 (38200)
  Cycle 1 Day 1 After Infusion: number analyzed (Participants) | 32 | 31 | 38
  Cycle 1 Day 1 After Infusion | 11900 (6410) | 9890 (4780) | 10800 (6230)
  Cycle 3 Day 1 Prior to Infusion: number analyzed (Participants) | 25 | 24 | 28
  Cycle 3 Day 1 Prior to Infusion | 238 (276) | 147 (60.9) | 161 (70.0)
  Cycle 3 Day 1 Before End of Infusion: number analyzed (Participants) | 22 | 23 | 27
  Cycle 3 Day 1 Before End of Infusion | 33800 (38600) | 23500 (21600) | 26800 (31900)
  Cycle 3 Day 1 After Infusion: number analyzed (Participants) | 23 | 23 | 28
  Cycle 3 Day 1 After Infusion | 20000 (30900) | 11200 (5160) | 14700 (14600)

ADVERSE EVENTS:
Time Frame: From the first study drug administration to the data cutoff date: 17 February 2021 (up to approximately 68 months).
Description: All-cause mortality is reported for deaths that occurred during the study based on the ITT population, which included all randomized participants. Serious and other adverse events were reported based on the safety population, which included all randomized participants who received at least one dose of any study medication.
Arm/Group | Arm C: Nab-Paclitaxel + Carboplatin | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin | Arm A: Atezolizumab + Paclitaxel + Carboplatin
All-Cause Mortality (participants affected / at risk) | 252/340 | 245/343 | 243/338
Serious Adverse Events (participants affected / at risk) | 96/334 | 168/334 | 151/332
Other Adverse Events (participants affected / at risk) | 315/334 | 325/334 | 315/332
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm C: Nab-Paclitaxel + Carboplatin (N=334) | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin (N=334) | Arm A: Atezolizumab + Paclitaxel + Carboplatin (N=332)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3) | 7 (7) | 6 (6)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 5 (5) | 13 (15) | 16 (16)
HAEMOLYSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 2 (2)
PANCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 3 (3) | 2 (3) | 6 (6)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 0 (0) | 5 (5)
ATRIAL THROMBOSIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
CARDIAC FAILURE (Cardiac disorders) | 1 (2) | 2 (2) | 1 (1)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2)
CARDIAC TAMPONADE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (2) | 1 (1)
TRACHEO-OESOPHAGEAL FISTULA (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 1 (1)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOPITUITARISM (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 4 (5) | 6 (6) | 3 (4)
DUODENAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
GASTROINTESTINAL NECROSIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL TOXICITY (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PANCREATITIS CHRONIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
ASTHENIA (General disorders) | 1 (2) | 0 (0) | 2 (2)
CHEST PAIN (General disorders) | 2 (2) | 0 (0) | 3 (5)
DEATH (General disorders) | 0 (0) | 8 (8) | 2 (2)
FATIGUE (General disorders) | 0 (0) | 3 (3) | 1 (1)
GAIT DISTURBANCE (General disorders) | 0 (0) | 0 (0) | 1 (1)
MALAISE (General disorders) | 1 (1) | 2 (2) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1)
OEDEMA (General disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1)
PERFORMANCE STATUS DECREASED (General disorders) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 5 (6) | 6 (6) | 6 (8)
AUTOIMMUNE HEPATITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
BILE DUCT STONE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (2)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATITIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
HEPATITIS TOXIC (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
IMMUNE-MEDIATED HEPATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
HAEMOPHAGOCYTIC LYMPHOHISTIOCYTOSIS (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 3 (3) | 6 (6)
CELLULITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
CHRONIC HEPATITIS C (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
COLONIC ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ENDOCARDITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
HEPATITIS B (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
INFECTED DERMAL CYST (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LUNG ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
MENINGITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PLEURAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 21 (21) | 33 (37) | 30 (32)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA HAEMOPHILUS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PSEUDOMONAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PULMONARY SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 2 (3) | 2 (3)
SEPSIS (Infections and infestations) | 6 (6) | 5 (5) | 10 (11)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
STOMATOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
URINARY TRACT INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
VASCULAR DEVICE INFECTION (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
CHEST INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
PERIORBITAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
RADIATION OESOPHAGITIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
RADIATION PNEUMONITIS (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
BLOOD LACTIC ACID INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
GENERAL PHYSICAL CONDITION ABNORMAL (Investigations) | 0 (0) | 0 (0) | 1 (2)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1) | 1 (1) | 3 (3)
PLATELET COUNT DECREASED (Investigations) | 2 (2) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 1 (1) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 4 (4)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
POLYMYOSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BENIGN SALIVARY GLAND NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
GALLBLADDER ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
INFECTED NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
TUMOUR EMBOLISM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BRAIN OEDEMA (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
EMBOLIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
EPILEPSY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
HEMIPLEGIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOTONIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
MOTOR DYSFUNCTION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
MYXOEDEMA COMA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DEVICE DISLOCATION (Product Issues) | 1 (1) | 0 (0) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
HALLUCINATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 4 (4) | 2 (2)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 2 (3) | 1 (1)
PROSTATITIS (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
BRONCHIAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (9) | 10 (14)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
DIAPHRAGMATIC PARALYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 7 (8) | 8 (8)
DYSPNOEA AT REST (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 6 (8)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
IMMUNE-MEDIATED PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
LARYNGEAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PARANASAL CYST (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (3)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 10 (10) | 10 (10)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 2 (2)
PNEUMOTHORAX SPONTANEOUS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 7 (7)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 3 (4)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
THERAPEUTIC EMBOLISATION (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
TRANSURETHRAL PROSTATECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
ARTERIAL STENOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
ARTERITIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
EMBOLISM (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMODYNAMIC INSTABILITY (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
SUPERIOR VENA CAVA SYNDROME (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm C: Nab-Paclitaxel + Carboplatin (N=334) | Arm B: Atezolizumab + Nab-Paclitaxel + Carboplatin (N=334) | Arm A: Atezolizumab + Paclitaxel + Carboplatin (N=332)
ANAEMIA (Blood and lymphatic system disorders) | 193 (244) | 188 (257) | 131 (153)
LEUKOPENIA (Blood and lymphatic system disorders) | 34 (54) | 42 (86) | 8 (8)
NEUTROPENIA (Blood and lymphatic system disorders) | 124 (214) | 121 (261) | 43 (61)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 92 (171) | 91 (163) | 46 (66)
HYPOTHYROIDISM (Endocrine disorders) | 2 (2) | 34 (40) | 27 (30)
ABDOMINAL PAIN (Gastrointestinal disorders) | 8 (8) | 9 (13) | 18 (20)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 17 (17) | 13 (17) | 12 (15)
CONSTIPATION (Gastrointestinal disorders) | 73 (85) | 101 (126) | 75 (94)
DIARRHOEA (Gastrointestinal disorders) | 77 (107) | 92 (135) | 94 (116)
NAUSEA (Gastrointestinal disorders) | 97 (137) | 131 (206) | 94 (139)
STOMATITIS (Gastrointestinal disorders) | 15 (17) | 22 (27) | 20 (24)
VOMITING (Gastrointestinal disorders) | 48 (59) | 67 (88) | 50 (64)
ASTHENIA (General disorders) | 66 (85) | 58 (81) | 77 (101)
CHEST PAIN (General disorders) | 18 (19) | 25 (31) | 28 (35)
FATIGUE (General disorders) | 88 (101) | 107 (137) | 97 (112)
MALAISE (General disorders) | 16 (24) | 18 (26) | 10 (14)
MUCOSAL INFLAMMATION (General disorders) | 9 (11) | 16 (23) | 17 (17)
OEDEMA PERIPHERAL (General disorders) | 22 (25) | 25 (32) | 23 (28)
PYREXIA (General disorders) | 34 (42) | 45 (66) | 46 (68)
NASOPHARYNGITIS (Infections and infestations) | 9 (11) | 21 (28) | 23 (35)
PNEUMONIA (Infections and infestations) | 16 (19) | 29 (30) | 23 (28)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 (6) | 10 (17) | 25 (38)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 (6) | 18 (24) | 18 (30)
URINARY TRACT INFECTION (Infections and infestations) | 16 (20) | 26 (45) | 18 (27)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 18 (23) | 40 (64) | 34 (56)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 17 (27) | 34 (64) | 31 (56)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 8 (8) | 17 (18) | 25 (33)
BLOOD CREATININE INCREASED (Investigations) | 3 (4) | 25 (28) | 16 (16)
NEUTROPHIL COUNT DECREASED (Investigations) | 65 (144) | 60 (132) | 18 (25)
PLATELET COUNT DECREASED (Investigations) | 59 (110) | 59 (128) | 40 (64)
WEIGHT DECREASED (Investigations) | 14 (14) | 32 (38) | 21 (22)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 36 (68) | 32 (64) | 12 (19)
DECREASED APPETITE (Metabolism and nutrition disorders) | 84 (98) | 82 (110) | 93 (109)
DEHYDRATION (Metabolism and nutrition disorders) | 11 (15) | 23 (33) | 20 (30)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 17 (19) | 18 (29) | 25 (28)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 23 (28) | 30 (39) | 24 (30)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 38 (56) | 54 (91) | 35 (47)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 5 (5) | 11 (17) | 17 (22)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 33 (37) | 53 (78) | 78 (107)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 16 (17) | 35 (40) | 33 (38)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 11 (14) | 23 (36)
MYALGIA (Musculoskeletal and connective tissue disorders) | 19 (24) | 22 (23) | 44 (63)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 17 (17) | 32 (35) | 35 (48)
DIZZINESS (Nervous system disorders) | 33 (42) | 32 (38) | 33 (35)
DYSGEUSIA (Nervous system disorders) | 22 (22) | 26 (30) | 15 (15)
HEADACHE (Nervous system disorders) | 18 (26) | 33 (40) | 38 (44)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 36 (39) | 34 (39) | 66 (73)
PARAESTHESIA (Nervous system disorders) | 15 (16) | 16 (17) | 28 (33)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 30 (35) | 48 (54) | 55 (68)
ANXIETY (Psychiatric disorders) | 10 (10) | 9 (10) | 17 (17)
INSOMNIA (Psychiatric disorders) | 27 (28) | 30 (34) | 29 (32)
COUGH (Respiratory, thoracic and mediastinal disorders) | 51 (61) | 65 (85) | 62 (69)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 19 (20) | 17 (17)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 57 (65) | 68 (100) | 64 (75)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 37 (43) | 34 (44) | 8 (9)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 18 (27) | 19 (29) | 18 (20)
ALOPECIA (Skin and subcutaneous tissue disorders) | 102 (103) | 114 (114) | 130 (134)
DRY SKIN (Skin and subcutaneous tissue disorders) | 5 (5) | 19 (21) | 13 (14)
PRURITUS (Skin and subcutaneous tissue disorders) | 13 (14) | 24 (36) | 32 (42)
RASH (Skin and subcutaneous tissue disorders) | 18 (19) | 47 (55) | 44 (57)
HYPOTENSION (Vascular disorders) | 12 (18) | 18 (25) | 22 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT02367794/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/94/NCT02367794/SAP_001.pdf